## STATISTICAL ANALYSIS PLAN

PROTOCOL NO: NCIG-007R

# Randomized, Double Blind, Placebo-Controlled Trial of the Efficacy of Intranasal Oxytocin for the Treatment of Alcohol Use Disorder

**Protocol Version No.:** 4.0 **Version Date:** 5 July 2022

#### **Study Sponsor:**

National Institute on Alcohol Abuse and Alcoholism

#### **Plan Authors:**

Charles B. Scott, Ph.D. Director of Biostatistics

Janet H. Ransom, Ph.D.
President
Fast-Track Drugs & Biologics, LLC
20010 Fisher Ave, Suite G
Poolesville, MD 20837

Daniel E. Falk, Ph.D.
Director of Biostatistics
Medications Development Branch
Division of Treatment Research
National Institute on Alcohol Abuse and Alcoholism
National Institutes of Health
6700B Rockledge Dr., Rm 1324
Bethesda MD 20892

**Version Number 1.0** 

Date: 7 September 2023

## STATISTICAL ANALYSIS PLAN

PROTOCOL NO: NCIG-007R

## Randomized, Double Blind, Placebo-Controlled Trial of the Efficacy of Intranasal Oxytocin for the Treatment of Alcohol Use Disorder

| Prepared by: | | Date: |
|--------------|-----------------------------------------|------------|
| - | Charles Scott, Ph.D. | |
| | Director of Biostatistics | |
| | Fast-Track Drugs & Biologics, LLC | |
| Reviewed by | <i>r</i> : | Date: |
| _ | Janet H. Ransom, Ph.D. | |
| | President | |
| | Fast-Track Drugs & Biologics, LLC | |
| Approved by | r: | Date: |
| | Daniel Falk, Ph.D. | |
| | Director of Biostatistics | |
| | Division of Treatment Research | |
| | National Institute on Alcohol Abuse and | Alcoholism |

| <i>2</i> . | INT | RODUCTION | 6 |
|---|---|---|---|
| 3. | PRO | OTOCOL SUMMARY | 7 |
| 3 | 3.1 | Study Objectives | 7 |
| | 3.1.1 | Primary | |
| | 3.1.2 | | |
| 3 | 3.2 | Study Design | 7 |
| 3 | 3.3 | Study Endpoints | |
| | 3.3.1 | Primary Efficacy Endpoint | |
| | 3.3.2 | Secondary Efficacy Endpoints | |
| | 3.3.3<br>3.3.4 | Exploratory Efficacy EndpointSafety Endpoints | |
| | 3.3.5 | Compliance | |
| 4.0 | | EFINITION OF ANALYSIS SETS | |
| 5.0 | | SSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS | |
| 4 | 5.1 | Alcohol Consumption Endpoints | |
| | 5.1.1 | Daily Quantity of Alcohol Consumption | 13 |
| | 5.1.2 | Drinking Days | |
| | 5.1.3 | Heavy Drinking Day | |
| | 5.1.4 | Days at Risk | 14 |
| | 5.1.5<br>5.1.6<br>Alcol | Weekly Percentage of Heavy Drinking Days and Weekly Percentage of Days Abstinent Percentage of Subjects with No Heavy Drinking Days and the Percentage of Subjects Abstine nol 14 | |
| | 5.1.7<br>5.1.8 | Weekly Mean Number of Drinks and Weekly Mean Number of Drinks per Drinking Day<br>World Health Organization Drinking Risk Categorical Scale | |
| 4 | 5.2 | Alcohol Use Disorder (MINI Version 7 – DSM5) | 15 |
| 4 | 5.3 | Barrett Impulsiveness Scale | 15 |
| 4 | 5.4 | Smoking and Cigarettes Smoked per Week | 16 |
| 4 | 5.5 | Nicotine use and Days of Other Nicotine Use per Week | 16 |
| | 5.6 | Experiences in Close Relationships – Relationship Structures Questionnaire (ECR- | -RS) 16 |
| 4 | 5.7 | Hyperkatifeia | 16 |
| 4 | 5.8 | Inventory of Drinking Situations (IDS-30) | 16 |
| 4 | 5.9 | PROMIS Questionnaires | 17 |
| | 5.9.1 | PROMIS – Alcohol-related Negative Consequences | 17 |
| | 5.9.2 | PROMIS – Sleep Disturbances | 17 |
| | 5.9.3 | PROMIS – Pain Interference | |
| 4 | 5.10 | Profile of Mood States (POMS) | |
| | 5.11 | Urge to Drink Scale (UDS) | |
| 6.0 | H | YPOTHESES TO BE TESTED | 18 |
| | 5.1 | Primary Efficacy Endpoint | 18 |
| | 5.2 | Secondary Efficacy Endnoints | 18 |

| <b>7.0</b> | SAMPLE SIZE CONSIDERATIONS | 19 |
|---|---|---|
| 8.0 | DATA QUALITY ASSURANCE | 19 |
| 9.0 | STATISTICAL CONSIDERATIONS | 20 |
| 9.1 | General Considerations | |
| 9.2 | Participant Accountability and Protocol Deviations | 20 |
| 9.3 | Demographics and Other Baseline Characteristics | 20 |
| 9.4 | Efficacy Analysis | 21 |
| | 4.1 Primary Analysis of Primary Efficacy Endpoint | |
| 9.4 | 4.2 Analysis of Secondary Endpoints | |
| 9.4 | 4.2.1 Secondary Drinking Endpoints | |
| 9.4 | 4.2.2 Alcohol Use and Craving Endpoints | |
| 9.4 | 4.2.3 Psychosocial Endpoints | 23 |
| 9.4 | 4.2.4 Nicotine-Related Endpoints | 23 |
| 9.4 | 4.3 Covariate Adjustment for the Analysis of Endpoints | 24 |
| 9.5 | Handling of Missing Data | 25 |
| 9.: | 5.1 Missing Data for Continuous Endpoints | |
| 9.6 | Safety Analysis | 25 |
| 9. | 6.1 Adverse Events | 25 |
| 9.0 | 6.2 Clinical Laboratory and Point of Care Tests | 26 |
| 9.0 | 6.3 Vital Signs, Weight, and ECG | 26 |
| | 6.5 CIWA-AR Scores | 26 |
| | 6.6 Buss-Perry Aggression Questionnaire (BPAQ) | 27 |
| | 6.7 Simplified Nutritional Appetite Questionnaire (SNAQ) | 27 |
| 9.0 | 6.8 University of Pennsylvania Smell Identification Test (UPSIT) | 27 |
| 9.7 | Drug Exposure and Retention | 27 |
| 9.8 | Analysis of Other Services Used | 28 |
| 9.9 | Concomitant Medications, Medical History, and Pregnancy Tests | 28 |
| 9.10 | Eligibility and Screen Failures | 28 |
| 9.11 | Exploratory Analyses | 28 |
| 9.12 | Ad hoc Analyses | 29 |
| <i>10</i> . | VALIDATION OF PROGRAMMING CODE | 29 |
| 11.0 | REFERENCES | |
| 12.0 | TABLE, LISTING, AND FIGURE SHELLS | 32 |

## 1. ABBREVIATIONS

| I. ABBKI | EVIATIONS |
|---|---|
| Abbreviation | Definition |
| AE | Adverse event |
| AICc | Akaike Information Criterion corrected for finite samples |
| AUC | Area under the concentration time curve |
| AUD | Alcohol Use Disorder |
| BAC | Blood alcohol concentration |
| BID | Twice daily |
| BIS | Barratt Impulsiveness Scale |
| BPAQ | Buss-Perry Aggression Questionnaire |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CIWA-AR | Clinical Institute Withdrawal Assessment for Alcohol-revised |
| CrCl | Creatinine clearance |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CTCAE | Common terminology criteria for adverse events |
| dL | Deciliter |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDMS | Electronic Data Management System |
| EOS | End of study |
| F | Fahrenheit |
| FA | Full Analysis |
| FDA | Food and Drug Administration |
| g | Gram |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transferase |
| hr | Hour |
| ICH | International Conference on Harmonization |
| IDS | Inventory of Drinking Situations |
| IRB | Institutional Review Board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| μg | Microgram |
| min | Minutes |
| MINI | MINI Neuropsychiatric Interview |
| mL | Milliliter |
| Mm | Millimeter |
| NHDD | No heavy drinking days |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| NIAAA | National Institutes on Alcohol Abuse and Alcoholism |
| Oz | Ounce |
| POMS | Profile of Mood State |
| PSNHDD | Percentage of subjects with no heavy drinking days |
| PT | Preferred term |
| RNA | Ribonucleic acid |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDU | Standard drinking unit |
| SNAQ | Simplified Nutritional Appetite Questionnaire |
| SOC | System Organ Class |
| STAI | Spielberger Trait Anxiety Inventory |
| THC | Tetrahydrocannabinol |
| TLFB | Timeline followback |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

#### 2. INTRODUCTION

This statistical analysis plan (SAP) for Protocol No. NCIG-007R, "Randomized, Double Blind, Placebo-Controlled Trial of the Efficacy of Intranasal Oxytocin for the Treatment of Alcohol Use Disorder" describes and expands upon the analytical plan presented in the protocol.

This document contains all planned analyses, reasons and justifications for these analyses for all study data. This plan also includes sample tables, figures, and listings that will be populated. The SAP will follow the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines as indicated in Topic E3 (Structure and Content of Clinical Study Reports), Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA) and ICH.

The following sources were used in preparation of this SAP:

- Protocol # NCIG-007R, Protocol Version No.: 4.0; Version Date: 05Jul2022
- ICH Guidance Topics E9, E3 and E8

#### 3. PROTOCOL SUMMARY

## 3.1 Study Objectives

#### **3.1.1 Primary**

The primary objective of the study is to compare the efficacy of intranasal oxytocin in reducing the weekly percentage of heavy drinking days over the 10 weeks of maintenance treatment among subjects with moderate to severe Alcohol Use Disorder (AUD). A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.

#### 3.1.2 Secondary

Secondary objectives include assessment of other measures of the effects of oxytocin compared with placebo on reduction of alcohol use as well as effects on alcohol craving, alcohol-related consequences, cigarette smoking and other nicotine use, psychological assessments, retention in the study, and safety and tolerability throughout the study.

## 3.2 Study Design

This study is a double-blind, randomized, placebo-controlled, parallel group, multi-site clinical trial designed to assess the efficacy of oxytocin compared with placebo to reduce drinking in 100 subjects (50 in each group) who report 4 or more Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition (DSM-5<sup>TM</sup>) symptoms of AUD. This study will be conducted at 4 clinical sites. If eligible for the study, subjects will be randomized using a stratified permuted block randomization procedure with "clinical site" as a stratification variable in an approximate 1:1 ratio (targeting 50 subjects per group) to receive either intranasal oxytocin or placebo for 12 weeks.

If eligible for the study, subjects will receive blinded intranasal oxytocin at 35 IU once per day or intranasal placebo (same volume once per day) for 2 weeks (initial tolerability assessment period), then for the next 10 weeks (maintenance period) subjects will receive oxytocin at 35 IU/twice per day (BID, totally daily dose 70 IU) or intranasal placebo (same volume twice per day)

Subjects will be seen in the clinic at screening visit(s), at randomization, and at Weeks 2, 3, 4, 6, 8, 10, and 13. During the alternate weeks when subjects will not be coming into the clinic (Weeks 5, 7, 9, 11, and 12), subjects will be contacted once during that week by telephone to encourage study drug compliance and to assess withdrawal, adverse events (AEs), and concomitant medication use. A final follow-up telephone interview will occur during Weeks 14/15 (1-to-2 weeks after the end of dosing).

Enrollment will be halted if 2 or more at least possibly related SAEs as judged by the investigator or medical monitor occur. If this occurs, a DSMB meeting will be convened and a decision, in conjunction with the study Sponsor, will be made regarding stopping the study.

The overall study schema is provided in Figure 1. The study schedule of visits and assessments is shown in Table 1.

Figure 1. Overview of Study Design



\*Telephone contact, otherwise visit is in clinic

Oxytocin for Alcohol Use Disorder Protocol Number: NCIG-007R

**Table 1. Schedule of Assessments** 

| | Screen | | | | | | ľ | Mainte | nance | | | | | <b>EOS</b> <sup>a</sup> | Safety<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | -2 to -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14/15 |
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | | 6 | | 7 | | 8 | | | 9 | |
| Informed Consent | X | | | | | | | | | | | | | | |
| Alcohol Breathalyzer | X | X | X | X | X | | X | | X | | X | | | X | |
| Urine Drug Screen <sup>b</sup> | X | X | X | X | X | | X | | X | | X | | | X | |
| Locator Form | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical/Surgical History | X | X <sup>c</sup> | | | | | | | | | | | | | |
| Physical Exam | $\mathbf{X}^{d}$ | X | X | X | X | | X | | X | | X | | | X | |
| MINI V 7.0.2 (AUD module at EOS) | X | | | | | | | | | | | | | X | |
| C-SSRS | | X | X | | | | X | | X | | X | | | X | |
| Clinical Chemistry <sup>e</sup> | X | | | | | | X | | X | | X | | | X | |
| Vital Signs | X | X | X | X | X | | X | | X | | X | | | X | |
| ECG (12-lead) | X | | | | | | | | | | | | | X | |
| Prior and Concomitant Meds | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CIWA-AR | X | X | X | X | X | | X | | X | | X | | | X | |
| Eligibility Checklist | X | X <sup>c</sup> | | | | | | | | | | | | | |
| Drug Compliance – Diary review | | X | X | X | X | | X | | X | | X | | | X | |
| Drug Accountability (vial weight) | | X | X | X | X | | X | | X | | X | | | X | |
| Pregnancy Test/Female Birth Control Methods | X | X | $\mathbf{X}^{\mathrm{f}}$ | | | | X | | X | | X | | | X | |
| Weight | X | | | | | | X | | X | | X | | | X | |
| Drinking Goal | X | | | | | | | | | | | | | | |
| AEs/SAEs | | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Other Services Used for Alcohol Use | | X | | | | | | | | | | | | X | |
| Problems <sup>g</sup> | | Λ | | | | | | | | | | | | A | |
| RANDOMIZATION | | X | | | | | | | | | | | | | |
| Brief Telephone Interview <sup>h</sup> | | | | | | X | | X | | X | | X | X | | |
| Take Control | | X | X | X | X | | X | | X | | X | | | | |
| Exit Interview | | | | | | | | | | | | | | X | |
| Treatment Referral | | | | | | | | | | | | | | X | |
| Follow-Up Telephone Interview | | | | | | | | | | | | | | | X |
| Final Subject Disposition | | | | | | | | | | | | | | | X |
| Subject Reported Outcomes | | | | | | | | | | | | | | | |

Statistical Analysis Plan: Protocol NCIG-007R, Version 1.0 Dated: 7 Sep 2023

Oxytocin for Alcohol Use Disorder Protocol Number: NCIG-007R

| | Screen | | | | Maintenance | | | | | | | <b>EOS</b> <sup>a</sup> | Safety<br>Follow-up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | -2 to -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14/15 |
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | | 6 | | 7 | | 8 | | | 9 | |
| Hyperkatifeia Scale | | X | | | | | | | | | | | | X | |
| Barrett Impulsivity Scale | | X | | | | | | | | | | | | | |
| Spielberger Trait Anxiety Inventory | | X | | | | | | | | | | | | | |
| BPAQ - SF <sup>i</sup> | | X | | | | | X | | X | | X | | | X | |
| Simplified Nutritional Appetite Questionnaire | | X | | | | | X | | X | | X | | | X | |
| Cigarette and other nicotine use | | X | | | | | X | | X | | X | | | X | |
| ECR-RS <sup>j</sup> | | X | | | | | X | | X | | X | | | X | |
| IDS-30 <sup>k</sup> | | X | | | | | | | | | | | | | |
| POMS | | X | | | | | X | | X | | X | | | X | |
| PROMIS – alcohol negative consequences | | X | | | | | X | | X | | X | | | X | |
| PROMIS – sleep disturbances | | X | | | | | X | | X | | X | | | X | |
| PROMIS – pain interference | | X | | | | | X | | X | | X | | | X | |
| UPSIT <sup>1</sup> | | X | | X | | | X | | X | | X | | | X | |
| Urge to drink questionnaire | | X | | | | | X | | X | | X | | | X | |
| Timeline followback (TLFB) | X | X | X | X | X | | X | | X | | X | | | X | |
| Brief Drinking Questionnaire <sup>m</sup> | | | | | | | | | | | | | | X | |

<sup>&</sup>lt;sup>a</sup> EOS=end of study. These assessments are to be done at Week 13 or if the subject discontinues early and agrees to a final clinic visit.

<sup>&</sup>lt;sup>b</sup> Test for opioids, cocaine, amphetamines, methamphetamine, THC, buprenorphine, methadone, benzodiazepines, oxycodone, 3,4-methylenedioxy-methamphetamine (MDMA), and barbiturates.

<sup>&</sup>lt;sup>c</sup> Updated prior to randomization.

<sup>&</sup>lt;sup>d</sup> Complete physical exam at screening including examination of the nares, plus examination of the nares at all other visits as indicated.

<sup>&</sup>lt;sup>e</sup> AST, ALT, total bilirubin, creatinine, sodium, and potassium.

f Only birth control methods are collected at this visit.

<sup>&</sup>lt;sup>g</sup> At baseline asks about lifetime treatment use and at EOS asks "since beginning this study"

<sup>&</sup>lt;sup>h</sup> AEs, concomitant medications, and drug compliance reminder.

<sup>&</sup>lt;sup>i</sup> Buss Perry Aggression Questionnaire – Short Form

<sup>&</sup>lt;sup>j</sup> Experiences in Close Relationships—Relationship Structures Questionnaire (ECR-RS) (attachment related anxiety)

<sup>&</sup>lt;sup>k</sup> Inventory of Drinking Situations

<sup>&</sup>lt;sup>1</sup> University of Pennsylvania Smell Identification Test

<sup>&</sup>lt;sup>m</sup>Only asked to subjects who request to withdraw from the study and are not willing to provide TLFB drinking data. This questionnaire will be asked at whatever constitutes the EOS visit.

#### 3.3 Study Endpoints

## 3.3.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the weekly percentage of heavy drinking days during the 10 week maintenance period (study weeks 3-12). A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.

#### 3.3.2 Secondary Efficacy Endpoints

Secondary endpoints that will be analyzed during the 10-week maintenance period (study weeks 3-12)include:

- 1. Percentage of subjects with no heavy drinking days during treatment
- 2. Percentage of subjects abstinent from alcohol during treatment
- 3. Percentage of subjects with a WHO drinking risk category decrease during treatment of:
  - a. At least 1-level
  - b. At least 2-levels
- 4. Endpoints analyzed monthly and with 1- and 2-month grace periods:
  - a. Percentage of subjects with no heavy drinking days during the period
  - b. Percentage of subjects abstinent from alcohol during the period
  - c. Percentage of subjects with WHO drinking risk category decrease during the period of:
    - at least 1 level
    - at least 2 levels
- 5. Percentage of days abstinent per week
- 6. Weekly mean number of drinks per week
- 7. Weekly mean drinks per drinking day
- 8. MINI AUD symptoms at end of study
- 9. Cigarettes smoked per week among smokers
- 10. Abstinence from cigarette smoking
- 11. Days used other nicotine products per week
- 12. Abstinence from nicotine use
- 13. Experiences in Close Relationships—Relationship Structures Questionnaire (ECR-RS) (attachment related anxiety)
- 14. PROMIS alcohol-related negative consequences
- 15. PROMIS sleep disturbances
- 16. PROMIS pain interference

- 17. Profile of Moods States (POMS) (including subscales)
- 18. Urge to Drink Scale (UDS)

## 3.3.3 Exploratory Efficacy Endpoint

Hyperkatifeia Scale score at end of study

### 3.3.4 Safety Endpoints

Safety endpoints will be analyzed over the entire treatment and follow-up period.

- 1. Vital signs
- 2. Physical examination of the nasal mucosa
- 3. Smell testing with the University of Pennsylvania Smell Identification Test (UPSIT)
- 4. Blood chemistries
- 5. Urine drug screen results
- 6. Blood alcohol concentration (BAC) by breathalyzer
- 7. AEs/SAEs
- 8. Electrocardiogram (ECG) results
- 9. Clinical Institute of Withdrawal Alcohol Revised (CIWA-AR) scores
- 10. Frequency of subjects with suicidal ideation at any time during the treatment period Columbia-Suicide Severity Rating Scale (C-SSRS)
- 11. Change in appetite Simplified Nutritional Appetite Questionnaire (SNAQ) scores and percentage of subjects with SNAQ scores ≤14.
- 12. Buss-Perry Aggression scores (BPAQ)

#### 3.3.5 Compliance

Compliance will be assessed using the Subject Diary and by weighing the used study drug vials prior to and after use to calculate the amount dispensed.

#### 4.0 DEFINITION OF ANALYSIS SETS

The study analysis populations will consist of the following:

**Full Analysis (FA) Set:** The full set is defined as subjects randomized to participate in the study who took at least one dose of investigational product. The full analysis set will be used to evaluate all efficacy and safety endpoints.

#### 5.0 ASSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS

## 5.1 Alcohol Consumption Endpoints

#### 5.1.1 Daily Quantity of Alcohol Consumption

Drinking will be assessed using the TLFB methodology (<u>Sobell et al., 1992</u>). The TLFB is a semi-structured interview that provides estimates of the daily quantity of alcohol consumption during specified time periods. It uses a calendar prompt and a number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drinking or other drug use during the target period. The procedure has been widely used in clinical and research contexts. It has demonstrated adequate levels of reliability and validity when administered as an in-person interview, over the telephone, and when administered via computer (<u>Carey 1997</u>; <u>Sobell et al., 1988</u>; <u>Sobell et al., 1996</u>).

After consent is signed, the TLFB interview will be performed for the 28-day period prior to signing consent. Thereafter, the interview will be for the previous days between the last assessment and the day prior to the day of the assessment.

If a subject requests to withdraw from the study but agrees to continued telephone contact to assess drinking, the TLFB will be performed over the phone for the duration of the study at a frequency acceptable to the study subject and site staff.

#### 5.1.2 Drinking Days

A drinking day is one calendar day in which the subject reported any alcohol consumption (i.e., > 0 standard drinking units [SDUs]). A standard drink contains approximately 0.6 fluid ounces (oz) of pure alcohol. The data given by the subjects on amount and type of alcoholic beverage(s) consumed will be converted to SDUs. An Excel spreadsheet customized for use in this study will be used for double data entry by clinical site staff to collect the TLFB drinking data. This spreadsheet contains a calculator to determine standard drink units (SDUs). Standard drink unit definitions are provided in Table 2.

#### **Table 2:** Standard Drink Unit Definitions

For Beer (~ 5% alcohol), the approximate number of SDUs in:

- 12 oz = 1.0
- 16 oz = 1.3
- 24 oz = 2.0
- 40 oz = 3.3

For malt liquor ( $\sim 7\%$  alcohol), the approximate number of SDUs in:

- 12 oz = 1.4
- 16 oz = 1.9
- 22 oz = 2.6
- 40 oz = 4.7

For table wine (~ 12% alcohol), the approximate number of SDUs in:

- 750 mL bottle = 25 oz = 5.0
- 5 oz glass = 1.0

#### • 10 oz glass = 2.0

For 80 proof spirits ( $\sim 40\%$  alcohol), or hard liquor, the approximate number of SDUs in:

- 1.5 oz (mixed drink) = 1.0
- 12.7 oz (pint) = 8.5
- 25 oz ( a fifth)= 17.0
- 1.75 L (59 oz) = 39.0

#### 5.1.3 Heavy Drinking Day

A heavy drinking day is defined as a day with 5 or more drinks (SDUs) for males and 4 or more drinks (SDUs) for females.

## 5.1.4 Days at Risk

If a subject is being treated at an inpatient facility, is incarcerated, or otherwise under confinement, each day spent in under these conditions is considered a reduction in the days at risk for drinking and is deducted from the denominator in calculations of rates of drinking days.

## 5.1.5 Weekly Percentage of Heavy Drinking Days and Weekly Percentage of Days Abstinent

Weekly percentage of heavy drinking days is the number of heavy drinking days in a 7-day period divided by 7 then multiplied by 100. The TLFB permits capturing data in a subsequent visit if a visit is missed; however, if fewer than 7 days are observed, then the denominator is the number of days observed in the 7-day period. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly percentage of days abstinent is similarly calculated by using the number of days abstinent instead of the number of heavy drinking days.

## 5.1.6 Percentage of Subjects with No Heavy Drinking Days and the Percentage of Subjects Abstinent from Alcohol

The percentage of subjects with no heavy drinking days is the number of subjects that have no heavy drinking days during the period of interest divided by the number of subjects with at least one day of non-missing drinking data during the period of interest, multiplied by 100.

The percentage of subjects abstinent from alcohol is calculated similarly, except the numerator is the number of subjects that have no drinking days during the period of interest.

## 5.1.7 Weekly Mean Number of Drinks and Weekly Mean Number of Drinks per Drinking Day

Weekly mean number of drinks is the sum of SDUs calculated to the tenths over 7 calendar days divided by the number of days with non-missing data. The quotient is multiplied by 7. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly mean number of drinks per drinking days utilizes the same numerator, and the denominator is the number of days with greater than 0 SDUs. Weeks where all days within the week are abstinent are assigned a value of 0 for weekly drinks per drinking day.

#### 5.1.8 World Health Organization Drinking Risk Categorical Scale

The WHO has developed a drinking risk categorical scale that can be used in a responder analysis approach to assess clinically relevant decreases in alcohol consumption (<u>Aubin et al., 2015</u>). Two dichotomous endpoints will be analyzed: WHO 1-level and WHO 2-level decrease in alcohol consumption. The WHO 1-level and 2-level decrease endpoints are the percentage of subjects experiencing at least a 1-level or 2-level decrease in WHO levels of alcohol consumption, respectively, from the level at baseline (the period including the 28 days before screening) to the level during period of interest. The WHO levels of average alcohol consumption per day are as follows:

| | Males | <b>Females</b> |
|----------------|------------|----------------|
| Low Risk | 1 to 40g | 1 to 20g |
| Medium Risk | 41 to 60g | 21 to 40g |
| High Risk | 61 to 100g | 41 to 60g |
| Very High Risk | 101+g | 61+g |

where 14g = 1 SDU (<u>WHO2000</u>). In computing the alcohol consumption level, average drinks per day will be used, computed as the sum of all drinking in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects will be included in a separate "Abstinent" category. A subject must have at least 1 week of data during a month to be considered non-missing.

## 5.2 Alcohol Use Disorder (MINI Version 7 – DSM5)

The AUD module of the MINI Neuropsychiatric Interview (MINI) specifies the severity of AUD into 3 categories based on the total number of symptoms to which the subject is coded "Yes" as follows:

Mild = 2 to 3 symptoms

Moderate = 4 to 5 symptoms

Severe = 6 or more symptoms

Subjects must have at least 4 symptoms to be eligible to participate in the study. The total number of symptoms being scored is 11. No imputation for missing values will be used.

## 5.3 Barrett Impulsiveness Scale

The Barratt Impulsiveness Scale (BIS) is a questionnaire designed to assess the personality/behavioral construct of impulsiveness. It is a 30-item scale with items scored on a 4-point scale (1=rarely/never; 2= occasionally; 3=often; 4=almost always/always). Items 1, 7, 8, 9, 10, 12, 13, 15, 20, 29, and 30 are reverse scored. The total score is the sum of the individual items. Separate subscale scores for Self-Control and Impulsive behavior will also be calculated. The BIS is among the baseline assessments that are performed only at Week 1.

## 5.4 Smoking and Cigarettes Smoked per Week

A quantity frequency interview at baseline and during treatment will include two questions to assess cigarette smoking behavior: 1) Over the past week, on how many days did you smoke cigarettes?; and 2) On the days you smoked during the past week, how many cigarettes did you smoke on average? At baseline subjects that answer "0" to question #1 are considered non-smokers for the study. Cigarettes per week is the answer to question #2 multiplied by the answer to question #1. No imputation for missing values will be used.

#### 5.5 Nicotine use and Days of Other Nicotine Use per Week

The cigarette smoking questionnaire will include a third question: 3) Over the past week, on how many days did you use other nicotine products (ex. chew, cigars, cigarillos, e-cigarettes, vape, gum, patch, etc...). A subject is positive for any nicotine use if the number of smoking days or the number of any other nicotine use days is greater than zero.

## 5.6 Experiences in Close Relationships – Relationship Structures Questionnaire (ECR-RS)

The Experiences in Close Relationships-Relationship Structures scale (<u>Farley et al, 2011</u>) is a questionnaire assessing two-dimensional relationship-specific attachment structures in adults beyond the traditional focus on romantic relationships. This is a 36-item questionnaire, of which only the first 18-item attachment-related anxiety scale will be assessed and evaluated. The presentation of the items were randomized on the form for subject completion. Each item is rated on a 7-point scale where 1 = strongly disagree and 7 = strongly agree. The attachment-related anxiety is determined by averaging the scores of these 18 items. However, items 9 and 11 are "reverse keyed".

## 5.7 Hyperkatifeia

Hyperkatifeia is defined as a greater intensity of negative emotional/motivational signs and symptoms during withdrawal from drugs of abuse in the withdrawal/negative affect stage of the addiction cycle (Koob 2021). Hyperkatifeia or negative emotional state is considered to be one of stages of addiction in the context of drug withdrawal (Koob and Le Moal 1997, Koob 2019). NIAAA has developed a 24-item self-report Hyperkatifeia Scale to capture negative emotionality after stopping alcohol drinking that will be assessed for the first time in this study of heavy drinkers with a diagnosis of moderate to severe AUD. The items address four measures associated with negative emotional state including anxiety, depression, stress, irritability and pain. Each item is is 5-point Likert scale assessing the intensity of the feelings and sensations experienced when not drinking alcohol. Higher scores are indicative of greater intensity of hyperkatifeia.

## 5.8 Inventory of Drinking Situations (IDS-30)

The IDS-30 is a 30-item patient completed questionnaire of reward and relief drinking that asks subjects to rate the frequency (0= never, 3 = almost always) of heavy drinking in various situations over the past year (Mann et al, 2018). Fifteen items measure reward drinking

tendencies and 15 items measure relief drinking tendencies. A subsequent evaluation of IDS-30 refined the definition of reward drinking to five items and relief drinking to five items (<u>Votaw et al</u>, 2022)

The reward drinking score is determined by summing the scores for these items: 6, 18, 21, 23, 27.

The relief drinking score is determined by summing the scores for these items: 9, 14, 15, 22, 25

Missing data is not imputed. All five questions within each scale must be answered for a score to be computed; otherwise, the scale is missing.

## 5.9 PROMIS Questionnaires

PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of personcentered measures that evaluates and monitors physical, mental, and social health in adults and children that were developed through the support of U. S. Department of Health and Human Services (https://www.healthmeasures.net/explore-measurement-systems/promis). Three of these assessments, described below, will be utilized in this study.

#### 5.9.1 PROMIS – Alcohol-related Negative Consequences

For negative consequences for alcohol use, the PROMIS Alcohol Negative Consequences – Short Form 7a questionnaire will be used to assess outcomes of alcohol use over the past 30 days. Each of the 7-items assesses the frequency of the negative alcohol-related consequence on 5-point Likert scale with higher scores indicating greater frequency. The scoring manual will be used to compute T-scores for each evaluation. All 7 questions must be answered for the form to be considered non-missing.

#### 5.9.2 PROMIS – Sleep Disturbances

For assessment of subject's sleep quality, the PROMIS Sleep Disturbance – Short Form 8b will be used. The questionnaire consists of 8 questions regarding the quality of sleep over the past 7 days. Each item on the measure is rated on a 5-point scale with a range of scores from 8 to 40 with higher scores indicating greater severity of sleep disturbance. The American Psychiatric Association has established levels of severity (none to slight [<55], mild [55.0 - 59.9], moderate [60 - 69.9] or severe [70 or higher] based on the T-score derived from a conversion table) {add reference to APA website|. At least 5 questions must be answered to be considered non-missing.

#### **5.9.3 PROMIS – Pain Interference**

For the assessment of pain interference, the shortened 8a version of the PROMIS for pain interference will be used to measure the self-reported consequences of pain over the past 7 days. This 8-item questionnaire assesses the degree to which pain interferes with various activities. Each item on the measure is rated on a 5-point scale with higher scores indicating greater pain

interference. The scale ranges from 8 to 40. The scoring manual will be used to compute T-scores for each evaluation. At least 5 questions must be answered to be considered non-missing.

## 5.10 Profile of Mood States (POMS)

The POMS measures dimensions of affect or mood (McNair and Heuchert 2005). It consists of 65 adjectives to which the subject responds according to a 5-point scale ranging from "not at all (0)" to "extremely (5)." Six subscale scores will be computed for items grouped as follows: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. A Total Mood Disturbance score will also be computed which consists of the sum of Tension-Anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, and Confusion-Bewilderment scores then subtracting the Vigor-Activity subscale score. A missing value within a subscale will be replaced by the average score of the answered items within the subscale; if 2 or more items within a subscale are missing then the entire subscale will be considered missing.

## 5.11 Urge to Drink Scale (UDS)

The UDS is a modified version of an assessment that was developed and validated by researchers at the University of Pennsylvania's Center for Studies of Addiction. This measure has been shown to be a valid and reliable instrument for assessing an individual's urge to drink alcohol. This scale has 5 items with 7 different responses to each item scored as 0 to 7. The questions pertain to the past week. The total score is the sum of the point scores for the individual items. Total scores of 10 or higher during treatment have been reported to be associated with increased risk for relapse. Missing values will not be imputed.

#### 6.0 HYPOTHESES TO BE TESTED

#### 6.1 Primary Efficacy Endpoint

It is hypothesized that oxytocin, as compared to placebo will reduce the weekly percentage of heavy drinking days over the 10-week maintenance period (study weeks 3-12). This hypothesis will be tested using other time periods during treatment.

## **6.2** Secondary Efficacy Endpoints

Over the 10-week maintenance period (study weeks 3-12), it is hypothesized that the oxytocin group, as compared to the placebo group, will:

- 1. Increase the percentage of subjects with no heavy drinking days
- 2. Increase the percentage of subjects abstinent from alcohol
- 3. Increase the percentage of subjects with a WHO drinking risk category decrease of:
  - a. 1-level
  - b. 2-levels
- 4. Increase the percentage of days abstinent per week

- 5. Decease the weekly mean number of drinks per week
- 6. Decrease the weekly mean drinks per drinking day
- 7. Decrease the number of MINI AUD symptoms
- 8. Decrease the cigarettes smoked per week among smokers
- 9. Increase the smoking abstinence rate among smokers
- 10. Decrease the weekly number of days of other nicotine use among other nicotine users
- 11. Increase the nicotine use abstinence rate among nicotine users (includes cigarettes)
- 12. Decrease in attachment related anxiety scores of the ECR-RS (attachment related anxiety)
- 13. Decrease in PROMIS sleep disturbance, alcohol-related negative consequences, and pain interference scores
- 14. Decrease in POMS subscales total mood disturbance, anger-hostility, fatigue-inertia, confusion-bewilderment, tension-anxiety and depression scores and/or increase vigor-activity
- 15. Decrease in the Urge to Drink scale scores

#### 7.0 SAMPLE SIZE CONSIDERATIONS

With an intake sample of 100 subjects (50 subjects per arm) and 12% attrition, it is projected that the sample size for primary endpoint analyses will be 88 (44 subjects per arm). The alpha level for the primary analyses will be 0.05, two-tailed. An estimate of the effect size (Cohen's d) for the investigational products is 0.60. Equal variances in both groups are assumed. These assumptions lead to a projected power of 0.80.

## 8.0 DATA QUALITY ASSURANCE

Data quality assurance will start with training of clinical investigative staff on data collection and assessment procedures including a Manual of Operations that describes what data to collect and procedures for completion of electronic case report form (eCRFs.) Completed eCRFs will be reviewed by Fast-Track Drugs and Biologics clinical monitors on a regular basis throughout the trial by comparison against the source documents.

All study data will come from the eCRFs and no other source data. eCRFs for this study were created using an electronic data management system (EDMS) based on Merge eClinicalOS. eCRFs were created using an established data dictionary for each variable including the field name, field type, field attributes, and coding for variables. Range checks, alpha-numeric requirements, and null/not null parameters were programmed as applicable. The back end database application is Oracle. Data entered into the EDMS system will be reviewed by Fast-Track clinical monitors and data managers. If incomplete or inaccurate data are found, the data will be queried in the system for site staff to address. The site will resolve data inconsistencies and errors using the EDMS with full audit trail of corrections being maintained within the

system. Corrections and changes to the data will be reviewed by Fast-Track clinical monitors and data managers.

Additional edit checks will be written to detect anomalies in the database. These checks will address inconsistencies (within visits, across visits), invalid/unusual values, missing values, and protocol violations. Edit checking will be validated on test data or actual clinical trial data. In addition to programmed edit checks, quality control examination of data will also be performed on reviews of data listings.

#### 9.0 STATISTICAL CONSIDERATIONS

#### 9.1 General Considerations

For descriptive purposes, dichotomous and categorical variables will be presented as number of observations and percentages; continuous variables will be given as means, standard deviations (SD), median, minimum (min) and maximum (max). Statistical tests will be two-tailed at a 0.05 Type I error rate. P-values for the primary and secondary endpoints of < 0.05 will be considered statistically significant. Endpoint data will also be screened for outliers and skewness. Appropriate non-parametric tests will be used to compare treatment groups on continuous baseline characteristics that are not normally distributed. Continuous endpoint data that are not normally distributed will be transformed using either a square root, logarithmic, or inverse transformation, the selection of which is determined by skewness and kurtosis statistics with values closest to zero and normalization of histograms. Cohen's d will be used to calculate the effect size for means. Odds ratios will be provided for all dichotomous outcomes. Descriptive statistics – mean, SD, median, min and max – of all endpoint data will be provided for each assessment point or summarized at each week for drinking endpoints. All data will be presented in listings. All analyses will be performed in the full analysis set.

## 9.2 Participant Accountability and Protocol Deviations

A summary will be prepared to show dropouts/retention over time in each group, along with the reason for early termination. The number of missing observations will be presented between groups. Protocol deviations will be presented as summaries by type of deviation.

## 9.3 Demographics and Other Baseline Characteristics

Summaries of the characteristics of the subjects in each of the study groups at baseline will be prepared for the full analysis set. Demographic characteristics (e.g., age, gender, race, and ethnicity) and other baseline characteristics including Barratt Impulsiveness scale (BIS), mood scales (e.g., Spielberger Trait Anxiety Inventory (STAI), Buss-Perry Aggression Questionnaire (BPAQ), POMS total and subscale scores), hyperkatifeia questionnaire, ECR-RS, Simplified Nutritional Appetite Questionnaire (SNAQ), PROMIS scales for alcohol negative consequences, sleep disturbances, and pain interference, University of Pennsylvania Smell Identification Test (UPSIT), and drinking goal) will be summarized by treatment group.

Baseline drinking parameters in the 28-days prior to the start of screening, age started drinking regularly, medical treatments for drinking in the past year, and other services used for alcohol problems in the past 4 weeks prior to consent will be summarized by treatment group. The

number and percentage of subjects with mild, moderate and severe symptoms of AUD and summary statistics for total number of symptoms will also be presented.

The numbers and percentages of subjects who are smokers, used any nictonine, used any other nicotine products, and any THC will be presented. The quantity of cigarettes smoked per week will be presented among smokers, and the number of days of other nicotine products used per week will be presented among subjects with any other nicotine product use.

Baseline drinking-associated consequences (CIWA-AR), alcohol craving (Urge to Drink Scale) total score, and Inventory of Drinking Situations (IDS) subscales of reward drinking and relief drinking will be summarized in a table.

Continuous variables will be summarized using means, standard deviations, medians, min, and max values. Categorical variables will be summarized using counts and percentages.

The comparability among the treatment groups with respect to the demographic and baseline variables will be evaluated by appropriate statistical methods. These will include t-tests for continuous variables, chi-square tests for categorical variables, and Fisher's exact test for binary variables. If a continuous variable is skewed, then the Wilcoxon rank sum test will be used on the raw data or a t-test on an appropriately transformed variable.

## 9.4 Efficacy Analysis

#### 9.4.1 Primary Analysis of Primary Efficacy Endpoint

The primary efficacy endpoint is the weekly percentage of heavy drinking days during the 10-week maintenance period (study weeks 3-12). The primary analysis of the primary endpoint will be a fully covaried, mixed-effect model for repeated measures employed on the Full Analysis Set (using an appropriate transformation of the endpoint, if needed; see Section 9.1). Treatment group, study week, treatment group by study week interaction, clinical site and baseline percentage of heavy drinking days will be covariates in the mixed effects model. The analyses will be performed using SAS PROC MIXED procedure Subjects are treated as a class variable and not continuous. The week, treatment group, and clinical site are also treated as class variables. Additional covariates may be selected using the method described in Section 9.4.3. The solution statement from SAS PROC MIXED is requested to provide the solution for the fixed effects parameters. A REPEATED statement specifies that values are repeated each week and subjects are nested within treatment group. The covariance structure is specified.

The selection of the covariance structure is performed using a simple repeated mixed effects model that includes treatment group as the only fixed effect and subject nested within treatment group as the only random effect. The covariance structure is selected from autoregressive, compound symmetry, Toeplitz, and unstructured. The Akaike Information Criterion (AICc) corrected for a finite sample is obtained from each of the four models for the four possible covariance structures to determine model fit. The smallest (minimum) AICc associated with one of the covariance structures is selected and the difference for each of the other three covariance structures is calculated. A graph is produced of the model fit statistics and relative difference for the four possible covariance structures.

If the primary endpoint requires a transformation, another mixed effect model that is identical to the primary analysis model will be run using the untransformed endpoint. Results based on the primary analysis model and the model of the untransformed endpoint will be presented in tabular form. The overall least squares means and least square means for each time point along with the 95% confidence intervals (CI) will be presented for the untransformed endpoint only (for descriptive purposes), while two-tailed p-values and Cohen's d will be presented for both the untransformed and transformed data. Inference and Cohen's d will be based upon the results using appropriately transformed data. A graph of the primary endpoint will be produced using the LSMEANs from the untransformed endpoint with p-values and Cohen's d comparing weekly differences obtained from the appropriately transformed variable.

Descriptive statistics will be reported for all study weeks (1-12) by treatment group.

#### 9.4.2 Analysis of Secondary Endpoints

Continuous secondary efficacy endpoints with repeated measures will also be analyzed based on data collected during the treatment period, including TLFB and other questionnaire data assessed at Week 13 that reflect data collected during this period.

In general, every continuous secondary efficacy endpoint with repeated measures is analyzed using a repeated measures mixed effects model as discussed in Section 9.4.1. Results will be presented using the same tabular and graphical formats detailed in Section 9.4.1. The primary analysis model is:

appropriately transformed endpoint = treatment + week + treatment\*week + clinical site + baseline equivalent of endpoint + other covariates (identified in Section 9.4.3).

It is anticipated that the covariance structure selected for the primary endpoint will also be used for secondary endpoints; however, the selection process detailed in Section 9.4.1 will be followed for each continuous secondary endpoint.

The primary analysis model for continuous endpoints measured at one time is a general linear model (GLM): appropriately transformed endpoint = treatment + clinical site + baseline equivalent of the endpoint + other covariates (identified in Section 9.4.3).

The primary analysis model for dichotomous endpoints is a logistic regression model that includes treatment + clinical site + other covariates (identified in Section 9.4.3). If fewer than 5 events are observed for a dichotomous endpoint then no logistic regression will be performed. In this situation Fisher's exact test will be used to compare treatment groups.

All analyses of secondary endpoints will use the Full Analysis Set.

Descriptive statistics of all secondary endpoints will be reported for all study weeks (1-12) or times at which they were measured within the treatment period, by treatment group.

#### 9.4.2.1 Secondary Drinking Endpoints

The continuous endpoints – percentage of days abstinent per week, weekly mean number of drinks per week, and weekly mean number of drinks per drinking day – will be analyzed using the mixed effects model specified in Section 9.4.2. Covariates for these models will be identified as in Section 9.4.3.

The dichotomous endpoints –percentage of subjects with a WHO 1-level decrease, and WHO 2-level decrease in alcohol consumption risk category, percentage of subjects with no heavy drinking days, and percentage of subjects abstinent from alcohol – will be assessed for the entire 10-week maintenance period, with 1- and 2-month grace periods, and Month 2 and Month 3. These endpoints will be analyzed with the logistic regression model specified in Section 9.4.2. Covariates for these models will be identified as in Section 9.4.3.

#### 9.4.2.2 Alcohol Use and Craving Endpoints

The MINI AUD module is assessed at screening and Week 13. The number of AUD symptoms at Week 13 is a continuous variable and will be modeled using a GLM specified in Section 9.4.2. Covariates for these models will be identified as in Section 9.4.3.

Craving is assessed using the Urge to Drink Scale which is assessed repeatedly during the treatment period. The total score will be analyzed using the mixed effect model approach detailed in Section 9.4.2. Covariates for this model will be identified as in Section 9.4.3.

#### 9.4.2.3 Psychosocial Endpoints

The POMS, ECR-RS, and the three PROMIS scales (including negative alcohol-related consequences, sleep disturbance, and pain interference) are continuous variables assessed repeatedly throughout the treatment period. The POMS includes the overall Total Mood Disturbance and other subscales, and each will be individually analyzed. The ECR-RS is a 36-item questionnaire of which only the first 18-item attachment-related anxiety scale will be assessed and analyzed. The three PROMIS scales employed in this study will be transformed into T-scores prior to analysis. The POMS, ECR-RS and PROMIS scores will be analyzed using the mixed effect model approach detailed in Section 9.4.2. Covariates for these models will be identified as in Section 9.4.3.

#### 9.4.2.4 Nicotine-Related Endpoints

The dichotomous endpoints – abstinence from smoking and abstinence from nicotine use – will be analyzed with the logistic regression model described in Section 9.4.2. Covariates for these models will be identified as in Section 9.4.3.

The mean number of cigarettes smoked in the past week is a continuous variable measured repeatedly during the treatment period. This endpoint will be analyzed only for those subjects who smoked at baseline. The data will be analyzed using the mixed effects described in Section 9.4.2. Covariates for this endpoint will be identified in Section 9.4.3.

The mean numbers of days of other nicotine product use is a continuous variable measured repeatedly during the treatment period. This endpoint will be analyzed only for those subjects who used other nicotine products at baseline. The data will be analyzed as described in Section 9.4.2. Covariates for this endpoint will be identified in Section 9.4.3.

#### 9.4.3 Covariate Adjustment for the Analysis of Endpoints

Covariates for the continuous efficacy endpoints measured repeatedly include the baseline equivalent of the endpoint, clinical site, treatment, time and the treatment by time interaction. Covariates for the continuous efficacy endpoints measured at a single time point include the baseline equivalent of the endpoint, clinical site, and treatment. Covariates for the dichotomous endpoints include treatment and clinical site; however, the number of covariates will depend upon the number of events. In general, 10 events per covariate are necessary for a stable logistic regression model (Peduzzi et al, 1996). If the number of events permits the inclusion of a baseline drinking covariate, the percentage of days abstinent will be used as the covariate for the percent subjects abstinent endpoint; the percentage of heavy drinking days will be used as the covariate for the percent subjects with no heavy drinking days endpoint; however, no baseline drinking covariate will be employed for the endpoint, percent subjects with a WHO decrease in alcohol consumption, as this endpoint already adjusts for baseline drinking in its calculation. If there are only 5-9 events in one of the dichotomous endpoints then a logistic regression will be performed with treatment group as the only covariate.

Clinical site is included as a covariate because it was chosen as a stratification variable to account for between site variability in outcome. Prior to conducting the logistic regression, a blinded analysis of site by treatment group by dichotomous secondary outcome will be performed to determine if every site has an outcome. Clinical sites with fewer than 3 events will be combined for the purpose of conducting the logistic regression. The baseline equivalent of the endpoint is a strong predictor of the endpoint and will generally be included as a covariate.

Additional covariates for the efficacy endpoints may include baseline characteristics with a theoretical and/or empirical basis for a relationship with a particular endpoint. Such characteristics may include, but are not limited to, drinking goal, age, and years of regular drinking (age minus age first started drinking alcohol regularly). Prior to the unblinding of the data, matrices of correlations between these baseline characteristics and each of the secondary efficacy endpoints, pooled across blinded treatment assignment, will be produced (using Pearson for continuous variables, Spearman for categorical outcomes). Selection of baseline variables to include as covariates in the models will be based on consideration of the following criteria: at least modest correlation with outcome (i.e.,  $r \ge 0.20$ ), and clinical expertise. Each endpoint may have a unique set of covariates. Care is taken to only select a limited number of covariates such that the models are not over fitted

## 9.5 Handling of Missing Data

## 9.5.1 Missing Data for Continuous Endpoints

Drinking data is collected in the TLFB. Prior to the subject dropping out of the study, every attempt will be made to continue to collect TLFB data. However, if the subject no longer wishes to participate in the collection of the TLFB, but agrees to a shorter drinking assessment using the Brief Drinking Questionnaire (BDQ), then, answers from the BDQ will be used in conjunction with the TLFB (if some TLFB data were provided by the subject) or in lieu of the TLFB (if no data were provided by the subject) to otherwise avoid missing data for drinking endpoints. Specifically, the BDQ has two questions assessing whether the subject had any heavy drinking days or drinking days during the period covered and will be used to assess the presence of a heavy drinking day or or a drinking day, respectively, for the drinking endpoints percentage of subjects with no heavy drinking days and percentage of subjects abstinent, respectively.

The primary analysis of the primary endpoint will be performed on available data in the Full Analysis Set with no imputation for missing data. However, a sensitivity analysis will be performed on the primary endpoint using multiple imputation for missing drinking data (<u>Jakobsen et al, 2017</u>). Multiple imputation replaces each missing value with a set of "m" plausible values that represent the uncertainty about the right value to impute. The multiple imputation method will be performed on transformed endpoint data, if a transformation is deemed necessary. The data will be evaluated for the pattern of missingness. If the data have monotone missingness then the regression method will be used. If the data have non-monotone missingness then the Monte Carlo method will be used (<u>Ratitch et al, 2013</u>). The imputation model will include a limited set of variables likely to be associated with missingness on the primary endpoint, excluding treatment assignment. The variables may include but are not limited to site, time and baseline alcohol use. The "m" imputed datasets each will be analyzed using mixed effects models then SAS PROC MIANALYZE will be used to combine the parameter estimates.

No imputation will be done for analysis of secondary endpoints.

#### 9.6 Safety Analysis

#### 9.6.1 Adverse Events

AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be grouped by system, organ, and class (SOC) and preferred term (PT) designation. The severity, frequency, and relationship of AEs to investigational product will be presented by SOC and PT groupings. Listings of each individual AE including start date, stop date, severity, relationship to IP, outcome, action taken (including any treatment administered), and duration will be provided.

Every AE will be assessed for whether or not it qualifies as an SAE. All SAEs will be categorized and listed according to the following categories: Congenital Anomaly or Birth Defect; Persistent or Significant Disability/Incapacity; Results in Death; Requires or Prolongs

Hospitalization; Other Medically Important Serious Event; or Life-Threatening. For deaths, the date and cause of death will be collected and listed. For hospitalizations, the dates of admission and release (discharge) will be collected and listed.

Each AE (based on PT) will be counted once only for a given study subject. If the same AE occurred on multiple occasions, the highest severity will be assumed. Thus, study subjects are not counted multiple times in a given numerator in the calculation of frequencies for a specific AE. C-SSRS reports of suicidality or suicidal ideation will be reported as AEs and analyzed as AEs if the investigator determines after an interview with the subject, that the responses are consistent with suicidal ideation or attempt. Tabulation of suicidal ideation by CSSRS will be presented without hypothesis testing; answers to the C-SSRS will be provided in a subject listing.

#### 9.6.2 Clinical Laboratory and Point of Care Tests

For clinical laboratory data, descriptive statistics will be generated for all tests performed at screening and at each clinic visit. If a laboratory analysis is repeated, the last measurement performed prior to the clinic visit will be used in the summary statistics for that clinic visit. If an unscheduled clinical laboratory visit occurs prior to a scheduled visit that is missed due to dropout, then the unscheduled visit will be used in the summary statistics for the missed scheduled clinical visit. If an unscheduled clinical laboratory visit occurs between two scheduled clinical visits, then the data from the unscheduled visit will only be presented in the listings and not in summary statistics. In addition, at each post-randomization clinic visit descriptive statistics for change from baseline will be generated. Laboratory values will be plotted as mean  $\pm$  standard error over time. All laboratory measurements will be presented in the listings.

Number and percentage of positive urine drug tests and pregnancy tests for screening visits and all treatment and follow-up visits will be tabulated. Results of all urine drug tests and pregnancy tests will be presented in the listings. The percentage of subjects with a positive urine drug test at any time post start of treatment will also be presented by test type and treatment group.

#### 9.6.3 Vital Signs, Weight, and ECG

Vital signs will be presented as summary statistics and change from baseline. The percentage of ECG results considered abnormal and clinically significant will be provided. Body weight will be presented as summary statistics and change from screening. No statistical tests will be performed. Vital signs, ECG results, and weight measurements for all visits will be presented in the listings.

#### 9.6.4 Blood Alcohol Concentration

The number and percent of subjects at any clinic visit that have a BAC > 0 will be tabulated. All BAC measurements will be presented in the listings.

#### 9.6.5 CIWA-AR Scores

The number and percentage of subjects who reported CIWA-AR scores  $\geq 10$  at any time after the start of dosing will be presented. Fisher's exact test will be performed. No modeling or imputation will be performed.

#### 9.6.6 Buss-Perry Aggression Questionnaire (BPAQ)

The short form version of the BPAQ is used in this study and is a 12-item self-report measure aggression. Each item is assessed on a 5-point Likert scale assessing the degree to which agreesion-related statements are characteristic of the subject during the past week. The BPAQ includes four subscales: physical aggression (4 items), verbal aggression (3 items), anger (2 items), and hostility (3 items) (Diamond and Magaletta, 2006). Scores for each subscale, which are the sum of the items, will be assessed individually. There is no total score for this scale.

Because the BPAQ is a repeated continuous measure, the BPAQ subscales wil be analyzed using the mixed effects described in Section 9.4.2. Descriptive statistics will be presented for each assessment by treatment group. No imputation will be performed.

#### 9.6.7 Simplified Nutritional Appetite Questionnaire (SNAQ)

The 8-item Council on Nutrition appetite questionnaire scale and its 4-item derivative The Simplified Nutritional Appetite Questionnaire (SNAQ) were developed to assess appetite and predict weight loss. The changes in appetite during the study will be evaluated using the clinically simpler version of the two scales, the SNAQ (Wilson 2005). The 4 item SNAQ asks: 1) My appetite is; 2) When I eat; 3: Food tastes; and 4) Normally I eat; with 5 possible responses that are scored numerically from 1 to 5. The sum of the responses is the total scale score. A SNAQ score ≤14 indicates significant risk of at least 5% weight loss within six months. The number and percentages of subjects in each group with a SNAQ score ≤14 at each visit will be summarized. Fisher's exact test will be used at each visit. No imputation for missing data will be performed. A mixed effects analysis on the continuous SNAQ score, as described in Section 9.4.2, will be used to evaluate change over time. No imputation will be performed.

#### 9.6.8 University of Pennsylvania Smell Identification Test (UPSIT)

The UPSIT will be assessed at screening and other clinic visits throughout the study to determine if intranasal investigational products cause any changes in sensory discrimination. It consists of 4 booklets each containing 10 microencapsulated (scratch and sniff) odors. The UPSIT test has been studied in individuals with alcohol addiction and has shown that this population generally had generally lower UPSIT scores that non-drinking controls. Outcomes will be captured in Adverse Event tables.

## 9.7 Drug Exposure and Retention

Medication compliance, defined as the amount of investigational product taken as a proportion of the total amount prescribed per protocol, will be evaluated for the oxytocin and placebo groups based on the Subject Diary. Average IU per day of investigational product taken based on the the vial weight difference prior to and after dispensment will also be reported overall and weekly will be reported for the oxytocin and placebo groups. Exposure and compliance averages will be compared across treatment groups using t-tests at each week and overall. If the data are meaningfully skewed then the Wilcoxon rank-sum test will be used. The same test will be used for each week and overall. The research participation rate, defined as percentage of subjects with complete drinking data, will be compared between treatment groups. A Fisher's Exact test will

be used for the overall participation rate, weekly tests will not be performed. In addition, the percentage of subjects discontinuing medication or early withdrawal from the study and a listing of these reasons for discontinuation will be provided. No statistical inference will be performed for reasons of discontinuation.

## 9.8 Analysis of Other Services Used

Weekly days of attendance at self-help meetings or other professional service providers to help reduce/quit drinking at study week 13 will be presented as summary statistics by treatment group. All other services used data will be presented in the listings.

## 9.9 Concomitant Medications, Medical History, and Pregnancy Tests

Concomitant and prior medications are collected at screening and at all study weeks and will be presented in a subject listing, as will pregnancy tests. Medical History will be coded using MedDRA, summarized in a table by treatment group and will be presented in subject listings. No statistical inference will be performed.

## 9.10 Eligibility and Screen Failures

Screen failures will be summarized in a table and provided in subject listings. Answers to eligibility criteria will be provided in the subject listings.

## 9.11 Exploratory Analyses

A number of variables will be tested as potential moderators of the medication treatment effect on the PHDD primary endpoint. Weeks 3-12 will be the period of interest. The model identified in Section 9.4.1 will be amended to include the potential moderator variable and the moderator by treatment group interaction. To aid with interpretation, continuous moderator variables will be dichotomized based on clinically accepted levels available from the literature. In the event a clinically meaningful cutoff is not available, LOESS curves will be used to identify a cut point. The LOESS curve analysis will use averaged PHDD data over study weeks 3-12, treatment group and the moderator of interest. In all approaches, an appropriate cutoff will be one that ensures a sufficient sample size in all resultant subgroups. The potential moderator variables are assessed at baseline and include: sex, IDS-30 reward/relief drinking, baseline drinks per week, measures of anxiety and depression (ECR-RS anxiety-related attachment, POMS subscales of depression and anxiety, Spielberger Trait Anxiety Inventory), Barratt Impulsiveness Scale, history of alcohol withdrawal (i.e., withdrawal question on the MINI for alcohol use disorder), and alcohol-related treatment goal.

There is interest in exploring the use of a new Hyperkatifeia Scale as an efficacy endpoint and moderator of drug response. Hyperkatifeia scores are assessed at Week 1 and Week 13 (EOS Visit 9). Exploratory analyses utilizing Hyperkatifeia Scale scores will include: 1) using the total score and subscales as an endpoints to assess treatment efficacy; and 2) conducting moderator analyses using total score and the subscales. The total score and subscales are the sum of the items.

## 9.12 Ad hoc Analyses

Ad hoc analyses may be performed on the Hyperkatifeia Scale as a planned part of exploring the utility of this scale including total scores, subscales, and individual items. Ad hoc analyses utilizing Hyperkatifeia Scale scores may include: 1) identification of baseline subsets and relationship to alcohol-related outcomes; 2) conducting mediator analyses; 3) factor analysis to better understand the underlying dimensions of hyperkatifeia; 4) validity of the Hyperkatifeia Scale by comparing to other measures (e.g., POMS and PROMIS scales or subscale scores); and 5) and further evaluation of the scales as endpoints to assess treatment efficacy. The data from this study could be used for meta-analyses with results of other studies to expand data availability for the proposed ad hoc analyses.

Ad hoc analyses may also be performed on the Drinking Goal questionnaire as a predictor and moderator of alcohol-related outcomes. Cutpoints for IDS-30 reward and relief drinkers have been proposed for high and low levels of each, creating 4 categories (Votaw et al, 2022). These categories will be related to drinking outcomes if there are sufficient sample sizes within each category.

#### 10. VALIDATION OF PROGRAMMING CODE

All SAS codes used to generate tables and listings will be validated and reviewed before being finalized. The validation process will be used to determine that the numbers are produced by a statistically valid method and that the execution of the computations is correct. Qualified personnel who have not previously been involved in the production of the original programming codes will perform the validation procedures. Methods of validation include independent programming and comparison to data listings. Tables will be reviewed for accuracy, consistency with this plan, consistency within tables, and consistency with corresponding output. Once validation is complete, a quality control reviewer will perform a final review of the documents for accuracy and consistency. Upon completion of validation and quality review procedures, all documentation will be collected and filed in the study documentation files at Fast-Track.

#### 11.0 REFERENCES

Aubin HJ, Reimer J, Nutt DJ, Bladstrom A, Torup L, Francois C, Chick J. Clinical relevance of as-needed treatment with nalmefene in alcohol dependent patients. Eur Addict Res. 2015;21:160–68

Carey KB. Reliability and validity of the time-line follow-back interview among psychiatric outpatients: a preliminary report. Psych Addic Behav. 1997;11, 26-33.

Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976:16:31-41.

Diamond PM, Magaletta PR. The short-form Buss-Perry aggression questionnaire (BPAQ-SF): A validation study with federal offenders. Assessment. 2006;13:227-240

Fraley RC, Heffernan ME, Vicary AM, and Brumbaugh C. The experiences in close relationships—relationship structures questionnaire: A method for assessing attachment orientations across relationships. Psychological Assessment. 2011;23:615-625.

Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162.

Koob GF, Le Moal M. Drug abuse: hedonic homeostatic dysregulation. Science. 1997. 278:52–58.

Koob GF. Neurobiology of opioid addiction: opponent process, hyperkatifeia, and negative reinforcement. Biol Psychiatry. 2019;87:44–53.

Koob GF. Drug Addiction: Hyperkatifeia/negative reinforcement as a framework for medications development. Pharmacol Rev. 2021;73:163-201.

Mann K, Roos CR, Hoffman S, Namovics H, Leménager T, Heinz A, Witkiewitz K. Precision medicine in alcohol dependence: A controlled trial testing pharmacotherapy response among reward and relief drinking phenotypes. Neuropsychopharmacology. 2018:1-9.

Morean ME, DeMartini KS, Leeman RF, Pearlson GD, Anticevic A, Krishnan-Sarin S, Krystal JH, O'Malley S. Psychometrically improved, abbreviated versions of three classic measures of impulsivity and self control. Psych Assess 2014;26:1003-1020.

McNair DM, Heuchert JWP. Profile of Mood States (POMS) Multi-Health Systems, Tonawanda, NY. 2005.

Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9.

Ratitch B, O'Kelly M, Tosiello R. Missing data in clinical trials: from clinical assumptions to statistical analysis using pattern mixture models. Pharm Stat. 2013 Nov-Dec;12(6):337-47.

Sobell LC, Sobell MB. Timeline followback: a technique for assessing self-reported alcohol consumption. In Litten, R. Z. and Allen, J.P. (Eds.) Measuring alcohol consumption: psychosocial and biochemical methods. Totowa, NJ: Humana Press (pp. 41-72) 1992.

Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988;83:393-402.

Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend 1996;42:49-54.

Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.

Votaw VR, Mann K, Kranzler HR, Roos CR, Nakovics H, Witkiewitz K. Examining a brief measure and observed cutoff scores to identify reward and relief drinking profiles: Psychometric properties and pharmacotherapy response. Drug Alcohol Depend. 2022 Mar 1;232:109257.

Wilson M-MG, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr 2005;82:1074–81.

World Health Organization (WHO): International Guide for Monitoring Alcohol Consumption and Related Harm. Geneva, WHO, 2000. Available at: http://whqlibdoc.who.int/hq/2000/who msd msb 00.4.pdf.

## 12.0 TABLE, LISTING, AND FIGURE SHELLS

| Table 1: | Subject Disposition - All Consented Subjects | 38 |
|---|---|---|
| Table 2: | Reasons for Screen Failure – All Consented Subjects | 39 |
| Table 3: | Exposure to Investigational Products Based on Subject Diary | 39 |
| Table 4: | Percent Compliance to Investigational Products Based on Subject Diary | |
| Table 5: | Exposure to Investigational Products Based on Weight of Vials | |
| Table 6: | Percent Compliance to Investigational Products Based on Weight of Vials | |
| Table 7: | Summary of Medical History | |
| Table 8:` | Exit Interview | 41 |
| Table 9: | Research Participation by Treatment Group and Week | 43 |
| Table 10: | Number and Percent of Subjects with Drinking Data Provided by the Brief Drin | king |
| Questionna | ire instead of the TLFB | |
| Table 11: | Demographic Characteristics | 45 |
| Table 12: | Baseline DSM-5 Disorders | 48 |
| Table 13: | Baseline Drinking-related Behavior and Characteristics | 49 |
| Table 14: | Baseline Drinking by TLFB | 51 |
| Table 15: | Baseline Other Substance Use | 53 |
| Table 16: | Baseline POMS | 54 |
| Table 17: | Baseline Alcohol-Related Craving, Consequences, and Withdrawal | 55 |
| Table 18: | Baseline Mood Questionnaires | 56 |
| Table 19: | Baseline ECR-RS | 58 |
| Table 20: | Baseline SNAQ | 58 |
| Table 21: | Baseline PROMIS Subscales | 59 |
| Table 22: | Baseline UPSIT | 60 |
| Table 23: | Weekly Percentage of Heavy Drinking Days from Baseline to Week 12 | 62 |
| Table 24: | Percentage of Heavy Drinking Days per Week -Mixed Effects, Weeks 3-12, No | ) |
| Imputation | 62 | |
| Table 25: P | ercentage of Heavy Drinking Days per Week – Multiple Imputation for Missing | |
| Values, Mix | ked Effects, Weeks 3-12 | |
| Table 26: | Drinks per Week from Baseline to Week 12 | 66 |
| Table 27: | Drinks per Week – Mixed Effects, Weeks 3-12 | |
| Table 28: | Drinks per Drinking Day from Baseline to Week 12 | 68 |
| Table 29: | Drinks per Drinking Day – Mixed Effects, Weeks 3-12 | 68 |
| Table 30: | Percent Days Abstinent from Baseline to Week 12 | 68 |
| Table 31: | Percent Days Abstinent – Mixed Effects, Weeks 3-12 | 68 |
| Table 32: | WHO Shift Baseline to Weeks 3-12 | |
| Table 33: | WHO 1-Level Decrease in Alcohol Consumption – Weeks 3-12 | 69 |
| Table 34: | WHO 1-Level Decrease in Alcohol Consumption – Full Model, Logistic | |
| Regression, | Weeks 3-12 | 70 |
| Table 35: | WHO 1-Level Decrease in Alcohol Consumption – Weeks 9-12 (2 Month Grace | |
| Table 36: | WHO 1-Level Decrease in Alcohol Consumption - Full Model, Logistic Regres | |
| Weeks 9-12 | 2 (2 Month Grace) | 70 |
| Table 37: | WHO 1-Level Decrease in Alcohol Consumption – Weeks 5-12 (1 Month Grace | e) 70 |
| Table 38: | WHO 1-Level Decrease in Alcohol Consumption - Full Model, Logistic Regres | sion, |
| Weeks 5-12 | 2 (1 Month Grace) | |

| Table 39: | WHO 1-Level Decrease in Alcohol Consumption Monthly | 1 |
|---|---|---|
| Table 40: | Monthly Summary of WHO 1-Level Decrease in Alcohol Consumption – Full | |
| Model | 71 | |
| Table 41: | WHO 2-Level Decrease in Alcohol Consumption – Weeks 3-12 | 2 |
| Table 42: | WHO 2-Level Decrease in Alcohol Consumption - Full Model, Logistic Regression | ı, |
| Weeks 3-12 | 72 | |
| Table 43: | WHO 2-Level Decrease in Alcohol Consumption – Weeks 9-12 (2 Month Grace) 72 | 2 |
| Table 44: | WHO 2-Level Decrease in Alcohol Consumption - Full Model, Logistic Regression | i, |
| Weeks 9-12 | (2 Month Grace) | 2 |
| Table 45: | WHO 2-Level Decrease in Alcohol Consumption – Weeks 5-12 (1 Month Grace) 72 | 2 |
| Table 46: | WHO 2-Level Decrease in Alcohol Consumption - Full Model, Logistic Regression | ١, |
| Weeks 5-12 | (1 Month Grace) | 2 |
| Table 47: | WHO 2-Level Decrease in Alcohol Consumption Monthly | 2 |
| Table 48: | Monthly Summary of WHO 2-Level Decrease in Alcohol Consumption – Full | |
| Model | 72 | |
| Table 49: | Subjects Abstinent from Alcohol – Weeks 3-12 | 3 |
| Table 50: | Subjects Abstinent from Alcohol - Full Model, Logistic Regression, Weeks 3-12.73 | 3 |
| Table 51: | Subjects Abstinent from Alcohol – Weeks 9-12 (2 Month Grace) | 3 |
| Table 52: | Subjects Abstinent from Alcohol - Full Model, Logistic Regression, Weeks 9-12 (2 | |
| Month Grac | e) | 3 |
| Table 53: | Subjects Abstinent from Alcohol – Weeks 5-12 (1 Month Grace) | 4 |
| Table 54: | Subjects Abstinent from Alcohol - Full Model, Logistic Regression, Weeks 5-12 (1 | |
| Month Grac | e) | 4 |
| Table 55: | Subjects Abstinent from Alcohol Monthly | 4 |
| Table 56: | Monthly Summary of Subjects Abstinent from Alcohol – Full Model | 4 |
| Table 57: | Subjects No Heavy Drinking Days – Weeks 3-12 | |
| Table 58: | Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 3-12 75 | |
| Table 59: | Subjects No Heavy Drinking Days – Weeks 9-12 (2 Month Grace) | 5 |
| Table 60: | Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 9-12 | |
| | race) | 6 |
| Table 61: | Subjects No Heavy Drinking Days – Weeks 5-12 (1 Month Grace) | |
| Table 62: | Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 5-12 | |
| | race) | 6 |
| Table 63: | Subjects No Heavy Drinking Days Monthly | |
| Table 64: | Monthly Summary of Subjects No Heavy Drinking Days – Full Model | |
| Table 65: | Urge to Drink Scale – Each Evaluation During Maintenance Period | |
| Table 66: | Urge to Drink Scale – Full Model, Mixed Effects, Weeks 6-13 | |
| Table 67: | ECR-RS (attachment related anxiety) – Each Evaluation During Maintenance Period | |
| | 78 | |
| Table 68: | ECR-RS Attachment-Related Anxiety - Full Model, Mixed Effects, Weeks 6-13 78 | 8 |
| Table 69: | POMS – Each Evaluation During Maintenance Period | |
| Table 70: | POMS Tension-Anxiety – Full Model, Mixed Effects, Weeks 6-13 | |
| Table 71: | POMS Depression-Dejection – Full Model, Mixed Effects, Weeks 6-13 80 | |
| Table 72: | POMS Anger-Hostility – Full Model, Mixed Effects, Weeks 6-13 | |
| Table 73: | POMS Vigor-Activity – Full Model, Mixed Effects, Weeks 6-13 | |

| Table 74: | POMS Fatigue-Inertia – Full Model, Mixed Effects, Weeks 6-13 | 80 |
|---|---|---|
| Table 75: | POMS Confusion-Bewilderment – Full Model, Mixed Effects, Weeks 6-13 | 80 |
| Table 76: | POMS Total Mood Disturbance – Full Model, Mixed Effects, Weeks 6-13 | 80 |
| Table 77: | PROMIS – Each Evaluation During Maintenance Period | 80 |
| Table 78: | PROMIS Alcohol Use Negative Consequences – Full Model, Mixed Effects, Wee | |
| 6-13 | 81 | |
| Table 79: | PROMIS Sleep Disturbances – Full Model, Mixed Effects, Weeks 6-13 | 81 |
| Table 80: | PROMIS Pain Interference – Full Model, Mixed Effects, Weeks 6-13 | 81 |
| Table 81: | Mean Cigarettes Smoked per Week (among smokers) – Each Evaluation During | |
| Maintenanc | e Period | 81 |
| Table 82: | Mean Cigarettes Smoked per Week (among Smokers) - Full Model, Mixed Effect | īS, |
| Weeks 6-13 | 82 | |
| Table 83: | Mean Days Use of Other Nicotine Products – Each Evaluation During Maintenand | ce |
| Period | 82 | |
| Table 84: | Mean Use of Other Nicotine Products – Full Model, Mixed Effects, Weeks 6-13 | 82 |
| Table 85: | Subjects Abstinent from Cigarettes among Smokers Weeks 6-13 | 82 |
| Table 86: | Subjects Abstinent from Cigarettes (among Smokers) – Logistic Regression, Weel | ks |
| 6-13 | 83 | |
| Table 87: | MINI AUD Number of Symptoms | 83 |
| Table 88: | MINI AUD Number of Symptoms – Analysis of Covariance, Week 13 | 83 |
| Table 89: | Overall Summary of Adverse Events | |
| Table 90: | Number and Percentage of Subjects with Adverse Events | 86 |
| Table 91: | Number and Percentage of Subjects with Adverse Events During Weeks 1 & 2 | 87 |
| Table 92: | Number and Percentage of Subjects with Adverse Events During Weeks 3-12 | |
| Table 93: | Summary of Subjects with Adverse Events by Severity and Relationship – Oxytoo | cin |
| | 87 | |
| Table 94: | Summary of Subjects with Adverse Events by Severity and Relationship – Placebe 87 | 0 |
| Table 95: | Number and Percentage of Subjects with Adverse Events by Maximum Severity | 88 |
| Table 96: | Number and Percentage of Subjects with Adverse Events by Maximum Severity | |
| | eks 1& 2 | 88 |
| Table 97: | Number and Percentage of Subjects with Adverse Events by Maximum Severity | |
| During Wee | · | 88 |
| Table 98: | Number and Percentage of Subjects with Adverse Events Occurring in >= 5% | 89 |
| Table 99: | Number and Percentage of Subjects with Adverse Events Leading to | |
| Discontinua | ation of Study | 89 |
| Table 100: | Number and Percentage of Subjects with Adverse Events Leading to | |
| Discontinua | ation of Study Medication | 90 |
| Table 101: | CIWA-AR Score > 10 at Least Once During Treatment | |
| Table 102: | Summary of Vital Signs and Body Weights | |
| Table 103: | Incidence of Abnormal Findings on Physical Exam in Nasal Mucosa | |
| Table 104: | Summary of Other Services Used During Treatment Period | |
| Table 105: | Summary of ECG Results | |
| Table 106: | Summary of Blood Chemistries | |
| Table 107: | Summary of Positive Urine Drug Tests, Pregnancy Test or BAC > 0.000 Any | |
| Time Durin | | 93 |

| Table 108: | BPAQ – Each Evaluation During Maintenance Period | 93 |
|---|---|---|
| Table 109: | BPAQ Physical Aggression Score Full Model, Mixed Effects, Entire | |
| Maintenanc | e Period | 94 |
| Table 110: | BPAQ Verbal Aggression Score Full Model, Mixed Effects, Entire | |
| Maintenanc | e Period | 95 |
| Table 111: | BPAQ Anger Score Full Model, Mixed Effects, Entire Maintenance Perio | d 95 |
| Table 112: | BPAQ Hostility Score Full Model, Mixed Effects, Entire Maintenance Per | riod95 |
| Table 113: | SNAQ – Untransformed, Each Evaluation During Maintenance Period | 96 |
| Table 114: | SNAQ Score < 14 at Each Visit During Treatment | 96 |
| Table 115: | SNAQ Total Score Full Model, Mixed Effects, Entire Maintenance Period | l 96 |
| Table 116: | Frequency of Subjects with Suicidal Ideation Any Time During the Study | 96 |
| Table 117: | Moderator: MINI AUD (Percent Heavy Drinking Days Weeks 3-12) | 98 |
| Table 118: | Moderator: POMS Tension-Anxiety (Percent Heavy Drinking Days Weeks 3 | |
| | 98 | , |
| Table 119: | Moderator: POMS Depression-Dejection (Percent Heavy Drinking Days We | eks |
| 3-12) | 99 | |
| Table 120: | Moderator: ECR-RS Attachment-Related Anxiety (Percent Heavy Drinking | Days |
| Weeks 3-12 | 2) 99 | 3 |
| Table 121: | Moderator: STAI (Percent Heavy Drinking Days Weeks 3-12) | 99 |
| Table 122: | Moderator: Drinking Goal (Percent Heavy Drinking Days Weeks 3-12) | 99 |
| Table 123: | Moderator: BIS Self Control (Percent Heavy Drinking Days Weeks 3-12) | |
| Table 124: | Moderator: BIS Impulsive Behavior (Percent Heavy Drinking Days Weeks 3 | 3-12) |
| | 99 | , |
| Table 125: | Moderator: Hyperkatifeia (Percent Heavy Drinking Days Weeks 3-12) | 99 |
| Table 126: | Hyperkatifeia Total Score | |
| Table 127: | Hyperkatifeia Total Score– Generalized Linear Model, Week 13 | 100 |
| Table 128: | Hyperkatifeia Stress/Anxiety Score | 100 |
| Table 129: | Hyperkatifeia Stress/Anxiety Score- Generalized Linear Model, Week 13 | |
| Table 130: | Hyperkatifeia Depression Score | 101 |
| Table 131: | Hyperkatifeia Depression Score- Generalized Linear Model, Week 13 | 101 |
| Table 132: | Hyperkatifeia Irritable Score | |
| Table 133: | Hyperkatifeia Irritable Score– Generalized Linear Model, Week 13 | 101 |
| Table 134: | Hyperkatifeia Pain Score | 101 |
| Table 135: | Hyperkatifeia Pain Score– Generalized Linear Model, Week 13 | 101 |
| Listing 1: | Subject Disposition - All Subjects | 103 |
| Listing 2: | Enrollment and Randomization – All Consented Subjects | 103 |
| Listing 3: | Reason not Eligible – Screen Failures | 104 |
| Listing 4: | Protocol Deviations | 104 |
| Listing 5: | Subjects Excluded from the Efficacy Analysis | 105 |
| Listing 6: | Demographics Data | 105 |
| Listing 7: | Baseline Drinking Characteristics. | |
| Listing 8: | MINI DSM5 Disorders | 107 |
| Listing 9: | MINI DSM5 AUD | 108 |
| Listing 10: | MINI AUD End of Study | 109 |
| Listing 11: | Medical History | 110 |

| Listing 12: | Surgical History | 111 |
|---|---|---|
| Listing 13: | Physical Exam | |
| Listing 14: | Drinking Treatment History | 112 |
| Listing 15: | Drinking Goal | 113 |
| Listing 16: | Daily and Weekly Standard Drink Units (TLFB) During Treatment | 114 |
| Listing 17: | Drinking Question. | |
| Listing 18: | Drinking Consequences, Craving, Appetite, and Anxiety | 114 |
| Listing 19: | UPSIT Scores | |
| Listing 20: | POMS Scores | |
| Listing 21: | PROMIS Scale Scores | 116 |
| Listing 22: | Smoking Data | |
| Listing 23: | Exit Interview | |
| Listing 24: | Other Services Use | 118 |
| Listing 25: | Drug Exposure | 119 |
| Listing 26: | Adverse Events | 120 |
| Listing 27: | Adverse Events Leading to Subject Discontinuation from Study | 121 |
| Listing 28: | Adverse Events Leading to Discontinuation of Investigational Product | 122 |
| Listing 29: | Serious Adverse Events | |
| Listing 30: | Columbia-Suicide Severity Scale | 124 |
| Listing 31: | BPAQ Scores | |
| Listing 32: | Blood Chemistries | 126 |
| Listing 33: | Pregnancy Test/Birth Control Data | 127 |
| Listing 34: | Blood Alcohol Concentration | 128 |
| Listing 35: | Urine Drug Screen | 128 |
| Listing 36: | Vital Signs and Body Weights | 129 |
| Listing 37: | Prior and Concomitant Medications | 129 |
| Figure 1: | Percent Heavy Drinking Days per Week Least Squares Means – Untransformed. | 130 |
| Figure 2: | Mean Drinks per Week Least Squares Means – Untransformed | 130 |
| | Mean Drinks per Drinking Day by Week Least Squares Means – Untransformed | |
| | Percentage of Subjects No Heavy Drinking Days Weeks 3-12 | |
| Figure 5: | Percentage of Subjects Abstinent Weeks 3-12 | 131 |
| Figure 6: | Percentage of Subjects with WHO 1-Level Decrease in Alcohol Consumption | |
| Weeks 3-12 | 131 | |
| Figure 7: | Percentage of Subjects with WHO 2-Level Decrease in Alcohol Consumption | |
| Weeks 3-12 | 131 | |
| Figure 8: | Cumulative Grace Periods for Percentage of Subjects No Heavy Drinking Days. | 132 |
| Figure 9: | Cumulative Grace Periods for Percentage of Subjects Abstinent | 132 |
| Figure 10: | Cumulative Grace Periods for Percentage WHO 1-Level Decrease in Alcohol | |
| Consumption | | |
| Figure 11: | Cumulative Grace Periods for Percentage WHO 2-Level Decrease in Alcohol | |
| Consumption | | |
| Figure 12: | Percentage Days Abstinent per Week Least Squares Means – Untransformed | 133 |
| Figure 13: | Weekly Number of Cigarettes Smoked in Smokers Least Squares Means – | |
| Untransform | | |
| Figure 14: | POMS Total Score Least Squares Means by Visit – Untransformed | 133 |
| Figure 15: | POMS Tension-Anxiety Least Squares Means by Visit – Untransformed | 133 |
|---|---|---|
| Figure 16: | POMS Depression-Dejection Least Squares Means by Visit – Untransformed. | 134 |
| Figure 17: | POMS Vigor-Activity Least Squares Means by Visit – Untransformed | 134 |
| Figure 18: | POMS Fatigue-Inertia Least Squares Means by Visit – Untransformed | 134 |
| Figure 19: | POMS Anger-Hostility Least Squares Means by Visit – Untransformed | 134 |
| Figure 20: | POMS Confusion-Bewilderment Least Squares Means by Visit – Untransform | ned |
| _ | 134 | |
| Figure 21: | PROMIS Alcohol Negative Consequences Least Squares Means by Visit – | |
| Untransformed | d | 134 |
| Figure 22: | PROMIS Sleep Disturbances Least Squares Means by Visit – Untransformed. | 134 |
| Figure 23: | PROMIS Pain Interference Least Squares Means by Visit – Untransformed | 134 |
| Figure 24: | ECR-RS Attachment-Related Anxiety Least Squares Means by Visit – | |
| Untransformed | <u>d</u> | 134 |
| Figure 25: | Clinical Chemistry Values Over Time | 135 |

## 12.1 Tables

# 12.1.1 Subject Disposition, Participation, Compliance

**Table 1:** Subject Disposition - All Consented Subjects

**Treatment Group** Placebo Oxytocin Total p-value<sup>1</sup> n (%) n (%) n (%) Number of Subjects Consented XXX Number of Subjects Screen Failed xxx(xx.x%)Number of Subjects Randomized XXX XXX XXXNumber of Subjects Randomized but Did Not Take Medication x (xx.x%) x (xx.x%) x(xx.x%)Number of Subjects Randomized and Took at Least One Dose of Study xx(xx.x%)xx(xx.x%)xxx(xx.x%)0.xxxMedication (Full Analysis Set) Number of Completed Subjects<sup>2</sup> xx(xx.x%)xx(xx.x%)xxx(xx.x%)0.xxxNumber of Subjects Discontinuing Medication, Remain in Study xx(xx.x%)xx(xx.x%)xx(xx.x%)0.xxxNumber of Subjects Discontinuing Medication, Drop out of Study xx(xx.x%)xx(xx.x%)xx(xx.x%)0.xxxReason for Discontinuation xx(xx.x%)xx(xx.x%)xx(xx.x%)Lost to follow up Died xx (xx.x%) xx (xx.x%) xx(xx.x%)xx(xx.x%)Adverse Event xx(xx.x%)xx(xx.x%)Logistical or practical reasons xx (xx.x%) xx (xx.x%) xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)Lack of perceived efficacy Absent from the protocol due to confinement in a controlled xx (xx.x%) xx(xx.x%)xx(xx.x%)environment Subject withdrew consent xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)Clinical deterioration xx(xx.x%)xx(xx.x%)xx(xx.x%)Prefer another treatment Protocol non-compliance xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)xx(xx.x%)Other reason

Programmer Notes: The discontinuation reasons are as given on the CRF. Include only the reasons actually used for the subjects in the study. If a subject discontinued, but the specific reason is missing, include 'Missing' as a row in the table. Use the order of discontinuation reasons as presented on the CRF page

<sup>&</sup>lt;sup>1</sup>p-value from Fisher's exact test for binary <sup>2</sup>Subjects completing Week 13 visit by phone or clinic

Table 2: Reasons for Screen Failure - All Consented Subjects

| Category | Reason | n (%) |
|-----------|----------------------------------|-------------|
| Inclusion | Too young | xxx (xx.x%) |
| | Refuse to take study medication | xxx (xx.x%) |
| Exclusion | Current substance abuse disorder | xxx (xx.x%) |
| | Other reason | xxx (xx.x%) |

Programmer list all reasons identified for screen failure with denominator being all consented subjects

Table 3: **Exposure to Investigational Products Based on Subject Diary** 

| | | | Plac | ebo | | | Oxytocin | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | N | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Insufflations <sup>2</sup> | | | | | | | | | | | | | |
| Week 1 (xx) <sup>3</sup> | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 2 (xx) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 3 (xx) Week 12 (xx) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Overall (Weeks 1-12) | | | | | | | | | | | | | |
| Total number of insufflations | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Total number of insufflations | XX | | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Weeks 1-2 | | XX.X | | | | | XX | XX.X | | | | | |
| Total number of insufflations | XX | | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Weeks 3-12 | | XX.X | | | | | XX | XX.X | | | | | |
| <sup>1</sup> p-value from t-test for continuous | variables | s (t) – skev | ved cont | inuous c | lata uses | the Wilc | oxon rai | nk-sum tes | t (w). | | | | |
| <sup>2</sup> Number of insufflations per week | | | | | | | | | | | | | |
| <sup>3</sup> xx maximum number.possibible in | week | | | | | | | | | | | | |

Table 4: Percent Compliance to Investigational Products Based on Subject Diary

| | | | Plac | ebo | | | | | Oxyt | ocin | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | n | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Insufflations <sup>2</sup> | | | | | | | | | | | | | |
| Week 1 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 2 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 3 Week 12 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Overall (Weeks 1-12) | | | | | | | | | | | | | |
| Total number of insufflations | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Total number of insufflations | XX | | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Weeks 1-2 | | XX.X | | | | | XX | XX.X | | | | | |
| Total number of insufflations | XX | | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Weeks 3-12 | | XX.X | | | | | XX | XX.X | | | | | |

<sup>&</sup>lt;sup>1</sup> p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w).
<sup>2</sup> percent is the # of sprays taken/#of sprays presecribed in a period

#### Table 5: **Exposure to Investigational Products Based on Weight of Vials**

Note that this is the same as Table 2 except using IU for dosing

#### Table 6: Percent Compliance to Investigational Products Based on Weight of Vials

Note that this is the same as Table 3 except using IU for dosing and percent is based upon IU taken/IU presecribed

**Table 7: Summary of Medical History** 

| MedDRA SOC/ | Placebo | Oxytocin |
|------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| SOC | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |

**Table 8:** Exit Interview

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| What medication do you believe you were taking? | | | | 0.xxx |
| Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | O.MM |
| Active | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Both Active & Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No Idea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other substance | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| Correctly Guessed Medication (Subjects that guessed a medicatio | n) | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | U.AAA |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | An (An,n/o) | Mit (Mil. M/V) | MA (MA,A70) | |
| Why did you answer above? | | | | 0.xxx |
| Had side effects | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Had no side effects | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Staff treated me different | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No improvement | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Had improvement | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Had a hunch | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| I just felt different | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| Do you feel the medication helped you to reduce drinking? | ( 0() | ( 0() | ( 0/) | 0.xxx |
| Very Much | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Much | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Moderately | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| A little | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not at all | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| How would you describe your experience taking the medication? | ? | , , | | 0.xxx |
| Experienced no unwanted side effects and benefited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced some unwanted side effects but benefited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced a lot unwanted side effects but benefited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced no unwanted side effects but did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced some unwanted side effects and did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced a lot of unwanted side effects and did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| If a friend were in need of help for a drinking problem, would yo | u recommend tak | ing the medication to | him/her? | 0.xxx |
| Yes, definitely | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | U.AAA |
| Yes, generally | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Neither yes nor no | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No, not really | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No, definitely not | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | Xx | XX | |
| f you were to need treatment in the future, would you choose to | | | | 0.xxx |
| Definitely yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Generally yes | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Neither yes or no | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No, not really | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Definitely not | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | Xx | XX | |
| How much do you think of yourself as wanting to please other po | <br> | er)? | | 0.xxx |
| More than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.7272 |
| Average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Less than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | Xx | XX | |
| 0 | | .1 ****1 | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c).

Table 9: Research Participation by Treatment Group and Week

| | | Placebo (N=x | x) | | Oxytocin (N=xx) | | |
|---|---|---|---|---|---|---|---|
| Study Week <sup>2</sup> | n | Cumulative n | Cumulative % | n | Cumulative n | Cumulative % | p-value <sup>1</sup> |
| Week 1 | XX | XX | xx.x% | XX | XX | XX.X% | 0.xxx |
| Week 2 | XX | XX | xx.x% | XX | XX | xx.x% | 0.xxx |
| Week 3 | XX | XX | XX.X% | XX | XX | XX.X% | 0.xxx |
| Week 4 | XX | XX | XX.X% | XX | XX | XX.X% | 0.xxx |
| Week 5 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 6 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 7 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 8 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 9 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 10 | XX | XX | xx.x% | XX | XX | xx.x% | 0.xxx |
| Week 11 | XX | XX | XX.X% | XX | XX | XX.X% | 0.xxx |
| Week 12 | XX | XX | XX.X% | XX | XX | XX.X% | 0.xxx |
| Week 13 | XX | XX | xx.x% | XX | XX | xx.x% | 0.xxx |

Fisher's exact test

Numbers and percentages are based on subjects that participated through a given week

Table 10: Number and Percent of Subjects with Drinking Data Provided by the Brief Drinking Questionnaire instead of the TLFB

| | J | Placebo | Ox | ytocin | |
|------------|----|---------|----|--------|----------------------|
| Study Week | n | % | n | % | p-value <sup>1</sup> |
| Week 3 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 4 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 5 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 6 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 7 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 8 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 9 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 10 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 11 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 12 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Overall | XX | xx.x% | XX | xx.x% | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Fisher's exact test

Note only rows with values above 0 will be presented

**Table 11:** Demographic Characteristics

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Age (years) | | ` | , , | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Gender at Birth | | | | 0.xxx |
| N | | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Race | | | | 0.xxx |
| N | XX | XX | XX | |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| African-American or Black | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| American Indian or Alaskan Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| More than one race or other race | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unknown or not reported | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | | | | 0.xxx |
| N | XX | XX | XX | |
| Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not reported | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unknown | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Race/Ethnicity | | | | 0.xxx |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Black | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Hispanic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Education (years) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Education | | | | 0.xxx |
| ≤ High School | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| > High School | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Marital Status | | | | 0.xxx |
| Legally Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | U.AAA |
| Living with Partner / Cohabitating | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Widowed | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Separated | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Divorced | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Never Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unknown | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | , , , | | | |
| Marital Status | | | | 0.xxx |
| Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Employment Pattern (last 30 days) | | | | 0.xxx |
| Full-time > 35 hrs /week | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.777 |
| Part-time regular | XX (XX.X%) | XX (XX.X%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) | |
| Part-time irregular | XX (XX.X%) | XX (XX.X%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) | |
| Student | xx (xx.x%) | XX (XX.X%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) | |
| Military Service | XX (XX.X%) | XX (XX.X%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) | |
| Unemployed | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | |
| Retired/Disabled | xx (xx.x%) | xx (xx.x%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) | |
| Homemaker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| In controlled environment | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | |
| Unknown | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Employment | | | | 0.xxx |
| Employed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Income | | | | 0.xxx |
| \$0-\$15,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$15,001-\$30,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$30,001-\$45,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$45,001-60,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$60,001-75,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$75,001-90,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$90,001-105,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$105,001-120,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| >\$120,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| Occupation | | | | 0.xxx |
| Corporate Executive or Major Professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Business Manager or Minor Professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Business Administrator, Small Business | | | | |
| Owner, or Semi-professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clerical Worker, Sales, or Technician | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Skilled Worker | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Semi-skilled Worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unskilled Worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other Occupation | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Unemployed (not paid for services) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Never Worked | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Missing/ Not Given | XX | XX | XX | |

<sup>1</sup> p-value from chi-square test (c), t-test for continuous data, and Fisher's exact test for binary categories (f)

**Table 12:** Baseline DSM-5 Disorders

| | Placebo | Oxytocin | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xxx) |
| DSM-5 Disorders <sup>1</sup> | | | , , |
| Major Depressive Episode | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Major Depressive Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidality | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicide Behavior Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Manic episode | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypomanic episode | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bipolar I Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bipolar II Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other Specified Bipolar Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Panic Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Agoraphobia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Social Anxiety Disorder (Social Phobia) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Obsessive Compulsive Disorder (Past month) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Posttraumatic Stress Disorder (Past month) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Alcohol Use Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Substance Abuse Disorder (Non-alcohol) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any Psychotic Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mood Disorder with Psychotic Features | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Major Depressive Disorder with Psychotic | | | |
| Features | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bipolar I Disorder with Psychotic Features | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anorexia Nervosa (past 3 months) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bulemia Nervosa (past 3 months) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Binge-eating Disorder (past 3 months) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Generalized Anxiety Disorder (past 6 months) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Medical, Organic, Drug Case Ruled Out | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Antisocial Personality Disorder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

As assessed by MINI

 Table 13:
 Baseline Drinking-related Behavior and Characteristics

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinking Goal (n, %) | | | | 0.xxx |
| Total Abstinence | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Reduce but not stop | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | | | | 0.xxx |
| Goal of no Heavy Alcohol Use (n, %) <sup>2</sup> | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Goal of at least 50% Reduction in Drinks Per | Week <sup>3</sup> | | | |
| N | xx | XX | XX | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Motivation to Reach Goal | | | | 0.xxx |
| N | xx | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx - xx) | |
| Confidence to Reach Goal | | | | |
| N | xx | XX | XX | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx - xx) | |
| AUD Symptom Severity | | | | 0.xxx |
| Moderate (4 or 5 symptoms) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Severe (6 or more symptoms) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| AUD Number of Symptoms | | | | 0.xxx |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 6 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| 7 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 8 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 9 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 10 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 11 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| AUD Number of Symptoms (continuous) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Age when first started drinking | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Lifetime Hospitalizations to<br>Reduce/Quit Drinking | xx | XX | xx | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | U.XXX |
| Median Median | XX XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Lifetime Hospitalizations for Illness/ | (лл-лл) | (лл-лл) | (\(\lambda - \lambda \lambda\) | |
| Injuries due to Drinking N | VV. | V.V | N.V. | 0.xxx |
| Mean (SD) | XX<br>XX.X (XX.XX) | XX<br>XX.X (XX.XX) | XX<br>XX.X (XX.XX) | U.XXX |
| Median (SD) | ` ′ | XX (XX.XX) | XX (XX.XX) | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Outpatient Visits to Reduce/Quit | (۸۸-۸۸) | (AA-AA) | (۸۸-۸۸) | |
| Drinking in Last 12 Months | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | J.11111 |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Lifetime Medical Detoxifications | () | ( 1) | (-1111) | |
| N | XX | XX | XX | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Past Year Number of Support Group Meetings <sup>4</sup> | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

Note: Percentages are based on the number of non-missing values in each variable.

**Table 14:** Baseline Drinking by TLFB

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Percentage of Heavy Drinking Days (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Percentage of Heavy Drinking Days (7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Percentage of Heavy Drinking Days (Percent Change Pre-screening Days -1 to -28 to 7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c) – Fisher's exact test for dichotomous variables (f)

<sup>&</sup>lt;sup>2</sup> No HDD and <=14 drinks per week for men or <=7 drinks per week women

<sup>&</sup>lt;sup>3</sup> Calculated using the subject's drinks per week during 28-day pre-screen period and the drinks per week obtained from the 7-day period on the Drinking Goal assessment

<sup>&</sup>lt;sup>4</sup> Examples include Alcoholics Anonymous (AA), 12 step, Save Ourselves, or similar group meetings attended for alcohol problems or drinking

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Week (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Drinks/Week (7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Drinks/Week (Percent Change Pre-screening Days -1 to -28 to 7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Drinks/Drinking Day (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Drinks/Drinking Day (7Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Drinks/Drinking Day (Percent Change Pre-screening Days -1 to -28 to 7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Percentage Days Abstinent (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Percentage Days Abstinent (7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx_ | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Percentage Days Abstinent (Percent Change Pre-screening Days -1 to - 28 to 7 Days Prior to Randomization) | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| WHO Risk Level | | | | 0.xxx |
| High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Very High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

**Baseline Other Substance Use Table 15:** 

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Cigarette Smoker? | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Any Nicotine Use? | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Any Other Nicotine Product Use? | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| THC | | | | 0.xxx |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable.

1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c)

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Cigarette Smoker? | | | | 0.xxx |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable. <sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical (c), Fisher's exact test for binary variables (f)

Programmer's note: Place the parenthesis and character after each p-value to denote the test

**Table 16:** Baseline POMS

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Tension-Anxiety | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Depression-Dejection | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Anger-Hostility | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Fatigue-Inertia | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Confusion-Bewilderment | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Vigor-Activity | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Total Mood Disturbance | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

Note: 1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

Table 17: Baseline Alcohol-Related Craving, Consequences, and Withdrawal

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| IDS Reward Drinking Score | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Scale Min-Max | | | (xx.x - xx.x) | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| IDS Relief Drinker Score | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| IDS Reward Drinker N (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| CIWA-AR | | | | 0.xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | XX.X | XX.X | XX.X | |
| (Min – Max) | (xx.x - xx.x) | (xx.x - xx.x) | (xx.x - xx.x) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| No. Subjects with Withdrawal Symptoms (CIWA ≥ 10) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |

Note: 1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w); chi-squared test for symptoms (c)

Programmer's note: Place the parenthesis and character after each p-value to denote the test

**Table 18:** Baseline Mood Questionnaires

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Scale | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| BIS Brief | | | | |
| Total Score | | | | |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | xxx.xx | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| STAI (T-Anxiety Scale) | | | | 0.xxx |
| N | XX | XX | XX | |

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Scale | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| BPAQ | | | | |
| Physical Aggression | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Anger | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Verbal Aggression | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Hostility | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

<sup>. &</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

**Table 19:** Baseline ECR-RS

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Subscale | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Attachment-related | | | | |
| Anxiety | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min - Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | · | (xx-xx) | |
| | | • | | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

**Table 20:** Baseline SNAQ

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| SNAQ | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| T 416 | | | | 0 |
| Total Score | | | | 0.xxx |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | |
| Median | XXX.XX | XXX.XX | XXX.XX | |
| (Min – Max) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Dichotomized | | | | 0.xxx |
| 15+ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| ≤14 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) Fisher's exact test for binary variables (f)

**Table 21:** Baseline PROMIS Subscales

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| Subscale | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Alcohol Use Negative Consequences | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD_ | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Sleep Disturbances | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD_ | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Pain Interference | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD_ | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| Median | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

**Table 22:** Baseline UPSIT

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| UPSIT | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Categories | | | | 0.xxx |
| Normosmia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Mild microsmia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Moderate microsmia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Severe microsmia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Anosmia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

## 12.1.2 Primary Efficacy Endpoint

Table 23: Weekly Percentage of Heavy Drinking Days from Baseline to Week 12

| | | Ox | ytocin | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean (SD) | Median | Min - Max | N | Mean (SD) | Median | Min - Max | p-value <sup>1</sup> |
| Baseline | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 1 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 2 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 3 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 4 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 5 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 6 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 7 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 8 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 9 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 10 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 11 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 12 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 3-12 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | |

<sup>&</sup>lt;sup>1</sup>t-tests for each individual week. Week 3-12 is evaluated in modeling

{programmer note: change test to Wilcoxon if the data are skewed}

Table 24: Percentage of Heavy Drinking Days per Week –Mixed Effects , Weeks 3-12, No Imputation

Type III Wald Tests<sup>1</sup>

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 10 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 9 | XXX | XXX.XX | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Values in Type III table are based upon transformed data {note to specify which transformation}

# Least Squares Means<sup>1</sup>

| | | | | 95% | ∕₀ CI | | | Untran | sformed | Trans | formed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

<sup>&</sup>lt;sup>1</sup>Values are based on untransformed data unless otherwise specified

Table 25: Percentage of Heavy Drinking Days per Week – Multiple Imputation for Missing Values, Mixed Effects, Weeks 3-12

**Least Squares Means** 

| | | | | 95% | % CI | | | Untran | sformed |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| Oxytocin | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

Statistical Analysis Plan: Protocol NCIG-007R, Version 1.0 Dated: 7 Sep 2023

## 12.1.3 Secondary Efficacy Endpoints

Table 26: Drinks per Week from Baseline to Week 12

| | | Ox | ytocin | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean (SD) | Median | Min - Max | N | Mean (SD) | Median | Min - Max | p-value <sup>1</sup> |
| Baseline | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 1 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 2 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 3 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 4 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 5 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 6 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 7 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 8 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 9 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 10 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 11 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 12 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | XXX |
| 3-12 | XX | xxx (xx.xx) | XXX | xxx - xxx | XXX | xxx (xx.xx) | XXX | xxx - xxx | |

<sup>&</sup>lt;sup>1</sup>t-tests for each individual week. Week 3-12 is evaluated in modeling

{programmer note: change test to Wilcoxon if the data are skewed}

Table 27: Drinks per Week – Mixed Effects, Weeks 3-12

Type III Wald Tests<sup>1</sup>

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 10 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 9 | XXX | XXX.XX | 0.xxx |

<sup>1</sup>Values in Type III table are based upon transformed data {note to specify which transformation}

## Least Squares Means<sup>1</sup>

| | | | | 95% | % CI | | | Untransformed | | Trans | formed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 4 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 5 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 11 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

| | | | | 95% CI | | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

<sup>&</sup>lt;sup>1</sup>Values are based on untransformed data unless otherwise specified

## Table 28: Drinks per Drinking Day from Baseline to Week 12

Same format as Table 18

## **Table 29:** Drinks per Drinking Day – Mixed Effects, Weeks 3-12

Same format as Table 19

## Table 30: Percent Days Abstinent from Baseline to Week 12

Same format as Table 18

## **Table 31:** Percent Days Abstinent – Mixed Effects, Weeks 3-12

Same format as Table 19

**Table 32:** WHO Shift Baseline to Weeks 3-12

| | Week 3-12 Category <sup>a</sup> | | | | |
|---|---|---|---|---|---|
| Baseline | Abstinent | Low Risk | Medium Risk | High Risk | Very High Risk |
| Category | n (%) | n (%) | n (%) | n (%) | n (%) |
| High Risk | | | | | |
| Very High Risk | | | | | |

<sup>&</sup>lt;sup>a</sup> Percent is based upon row denominator (eg # subjects with High Risk at baseline)

Same table for Oxytocin subjects only

Same table for Placebo subjects only

**Table 33:** WHO 1-Level Decrease in Alcohol Consumption – Weeks 3-12

| | Placebo | Oxytocin | Total |
|----------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| WHO 1-Level Decrease | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 34: WHO 1-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 3-12

| | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard Error | Wald Chi-Square | Pr > Chi-Square | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | |
| Treatment | Oxytocin | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

**Table 35:** WHO 1-Level Decrease in Alcohol Consumption – Weeks 9-12 (2 Month Grace)

Same style as Table 33

Table 36: WHO 1-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 9-12 (2 Month Grace)

Same style as Table 34

Table 37: WHO 1-Level Decrease in Alcohol Consumption – Weeks 5-12 (1 Month Grace)

Same style as Table 33

Table 38: WHO 1-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 5-12 (1 Month Grace)

Same style as Table 34

**Table 39: WHO 1-Level Decrease in Alcohol Consumption Monthly** 

| | Placebo | Oxytocin | Total |
|---------------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| Mo 2 WHO 1-Level Decrease | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mo 3 WHO 1-Level Decrease | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 40: Monthly Summary of WHO 1-Level Decrease in Alcohol Consumption – Full Model

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Model<br>Month <sup>a</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | OR | Upper CI | Lower CI |
| 2 | Treatment | Oxytocin | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 | Treatment | Oxytocin | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

## **Adjusted Prevalence Estimates**<sup>1</sup>

| | | | | | OR 95% CI | | |
|----------|-------|----------|-------|-------|-----------|----------|---------|
| Arm | Month | Estimate | SE | OR | Lower CI | Upper CI | p-value |
| Oxytocin | 2 | XX.XX | 0.xxx | 0.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | | | |
| Oxytocin | 3 | XX.XX | 0.xxx | 0.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | | | |

<sup>&</sup>lt;sup>1</sup>The adjusted prevalence rates are obtained from the monthly logistic regression models

Table 41: WHO 2-Level Decrease in Alcohol Consumption – Weeks 3-12

Same as Table 33

Table 42: WHO 2-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 3-12

Same as Table 34

**Table 43:** WHO 2-Level Decrease in Alcohol Consumption – Weeks 9-12 (2 Month Grace)

Same style as Table 33

Table 44: WHO 2-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 9-12 (2 Month Grace)

Same style as Table 34

**Table 45:** WHO 2-Level Decrease in Alcohol Consumption – Weeks 5-12 (1 Month Grace)

Same style as Table 33

Table 46: WHO 2-Level Decrease in Alcohol Consumption – Full Model, Logistic Regression, Weeks 5-12 (1 Month Grace)

Same style as Table 34

**Table 47: WHO 2-Level Decrease in Alcohol Consumption Monthly** 

Same style as Table 39

Table 48: Monthly Summary of WHO 2-Level Decrease in Alcohol Consumption – Full Model

Same style as Table 40
**Table 49:** Subjects Abstinent from Alcohol – Weeks 3-12

| Placebo | Oxytocin | Total |
|------------|----------------------|--------------------------------------|
| (N=xx) | (N=xx) | (N=xxx) |
| xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | (N=xx)<br>xx (xx.x%) | (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) |

Table 50: Subjects Abstinent from Alcohol – Full Model, Logistic Regression, Weeks 3-12

| | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | |
| Treatment | Oxytocin | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | |
| Site | 1 | х | XX.XXX | xx.xxx | XX.XXX | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

Table 51: Subjects Abstinent from Alcohol – Weeks 9-12 (2 Month Grace)

Same as Table 49

Table 52: Subjects Abstinent from Alcohol – Full Model, Logistic Regression, Weeks 9-12 (2 Month Grace)

## **Table 53:** Subjects Abstinent from Alcohol – Weeks 5-12 (1 Month Grace)

Same as Table 49

### Table 54: Subjects Abstinent from Alcohol – Full Model, Logistic Regression, Weeks 5-12 (1 Month Grace)

**Table 55:** Subjects Abstinent from Alcohol Monthly

| | Placebo | Oxytocin | Total |
|--------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| · | | | |
| Mo 2 Drinking Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mo 3 Drinking Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 56: Monthly Summary of Subjects Abstinent from Alcohol – Full Model

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Model<br>Month <sup>a</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | OR | Upper CI | Lower CI |
| 2 | Treatment | Oxytocin | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | xx.xxx |
| 3 | Treatment | Oxytocin | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup> Separate models are created for each month; only the treatment arm results are presented in the summary table

## **Adjusted Prevalence Estimates**<sup>1</sup>

| | | | | | OR 9 | 5% CI | |
|---|---|---|---|---|---|---|---|
| Arm | Month | Estimate | SE | OR | Lower CI Upper CI | | p-value |
| Oxytocin | 2 | XX.XX | 0.xxx | 0.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | | | |
| Oxytocin | 3 | XX.XX | 0.xxx | 0.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | | | |

<sup>&</sup>lt;sup>1</sup>The adjusted prevalence rates are obtained from the monthly logistic regression models

**Table 57:** Subjects No Heavy Drinking Days – Weeks 3-12

| | Placebo<br>(N=xx) | Oxytocin<br>(N=xx) | Total (N=xxx) |
|---|---|---|---|
| No Heavy Drinking<br>Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

 Table 58:
 Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 3-12

Same as Table 50

**Table 59:** Subjects No Heavy Drinking Days – Weeks 9-12 (2 Month Grace)

Table 60: Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 9-12 (2 Month Grace)

Sam as Table 50

**Table 61:** Subjects No Heavy Drinking Days – Weeks 5-12 (1 Month Grace)

Same as Table 49

Table 62: Subjects No Heavy Drinking Days – Full Model, Logistic Regression, Weeks 5-12 (1 Month Grace)

Same as Table 50

**Table 63:** Subjects No Heavy Drinking Days -- Monthly

Same style as Table 55

Table 64: Monthly Summary of Subjects No Heavy Drinking Days – Full Model

Same style as Table 56

**Table 65:** Urge to Drink Scale – Each Evaluation During Maintenance Period

| | | | 0 | xytocin | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 66: Urge to Drink Scale – Full Model, Mixed Effects, Weeks 6-13

Type III Wald Tests<sup>1</sup>

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|------------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | ARM*Week 3 | | XXX.XX | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Values in Type III table are based upon transformed data {note to specify which transformation}

### **Least Squares Means**

| | | | | 95% | % CI | | | Untran | sformed | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 13 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 13 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 67: ECR-RS (attachment related anxiety) – Each Evaluation During Maintenance Period

| | | | 0 | xytocin | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Anxiety | | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 68: ECR-RS Attachment-Related Anxiety – Full Model, Mixed Effects, Weeks 6-13

**Table 69:** POMS – Each Evaluation During Maintenance Period

| | | | O | xytocin | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Tension-Anxiet | y | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Depression-De | iection | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 13 | XX | XXX | XXX | XXX | | | XXX | XXX | XXX | XXX | XXX | XXX |
| Anger-Hostility | λλ | AAA | λλλ | AAA | XXX | XXX | XXX | AAA | λλλ | AAA | XXX | XXX |
| Baseline | 7/3/ | VVV | vvv | NWW. | VVV | VVV | WWW | WWW. | 777 | NWW. | WWW | WWW |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| _ | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Vigor-Activity | · I | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Fatigue-Inertia | | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Confusion-Bewi | ilderment | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Total Mood Dis | turbance | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 70: POMS Tension-Anxiety – Full Model, Mixed Effects, Weeks 6-13

Shell is the same style as Table 66

Table 71: POMS Depression-Dejection – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

Table 72: POMS Anger-Hostility – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

Table 73: POMS Vigor-Activity – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

Table 74: POMS Fatigue-Inertia – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

Table 75: POMS Confusion-Bewilderment – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

Table 76: POMS Total Mood Disturbance – Full Model, Mixed Effects, Weeks 6-13

Shell is same style as Table 66

**Table 77: PROMIS – Each Evaluation During Maintenance Period** 

| | | | 0 | xytocin | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Alcohol Negativ | ve Conseq | quences | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sleep Disturbar | nces | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Pain Interferen | ce | | | | | | | | | | | |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 78: PROMIS Alcohol Use Negative Consequences – Full Model, Mixed Effects, Weeks 6-13

Shell is the same style as Table 66

Table 79: PROMIS Sleep Disturbances – Full Model, Mixed Effects, Weeks 6-13

Shell is the same style as Table 66

Table 80: PROMIS Pain Interference – Full Model, Mixed Effects, Weeks 6-13

Shell is the same style as Table 66

Table 81: Mean Cigarettes Smoked per Week (among smokers) – Each Evaluation During Maintenance Period

| | | | 0 | xytocin | | | | | Pla | cebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 82: Mean Cigarettes Smoked per Week (among Smokers) – Full Model, Mixed Effects, Weeks 6-13
Same as Table 66

Table 83: Mean Days Use of Other Nicotine Products – Each Evaluation During Maintenance Period

Same as Table 81

**Table 84:** Mean Use of Other Nicotine Products – Full Model, Mixed Effects, Weeks 6-13 Same as Table 66

Table 85: Subjects Abstinent from Cigarettes among Smokers Weeks 6-13

| | Placebo | Oxytocin | Total |
|-----------------------------|------------|------------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| <b>Completely Abstinent</b> | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 86: Subjects Abstinent from Cigarettes (among Smokers) – Logistic Regression, Weeks 6-13

| | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | |
| Treatment | Oxytocin | х | XX.XXX | xx.xxx | XX.XXX | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | Overall | х | XX.XXX | xx.xxx | XX.XXX | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | 1 | х | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | |
| Site | 210 | х | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | |
| Cov | | х | XX.XXX | xx.xxx | xx.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |

**Table 87:** MINI AUD Number of Symptoms

| | | Oxytocin | | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 88: MINI AUD Number of Symptoms – Analysis of Covariance, Week 13

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | xxx | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| MINI AUD | 1 | xxx | XXX.XX | 0.xxx |

# **Least Squares Means**

| | | | 95% | 6 CI | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | xx.xxx | 0.xxx | XX.XXX |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

## 12.1.4 Safety Analyses

**Table 89:** Overall Summary of Adverse Events

| | Placebo | Oxytocin | Total | |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Number of AEs | XX | XX | XX | |
| Number of SAEs | XX | XX | XX | |
| Number (%) of subjects with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number (%) of subjects with at least one SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number (%) of subjects with at least one AE related <sup>2</sup> to study product | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number of AEs by severity | | | | |
| Mild | XX | XX | XX | |
| Moderate | XX | XX | XX | |
| Severe | XX | XX | XX | |
| Life-threatening | XX | XX | XX | |
| Number of AEs by relationship to study product | | | | |
| At least possibly related | XX | XX | XX | |
| Unrelated | XX | XX | XX | |
| Number of AEs by SAE status | | | | |
| No | XX | XX | XX | |
| Yes | XX | XX | XX | |

<sup>&</sup>lt;sup>1</sup>p-value from chi-square test <sup>2</sup> Related is possible, probable, or definite

**Table 90:** Number and Percentage of Subjects with Adverse Events

| MedDRA System Organ Class/ | Placebo | Oxytocin | p-value <sup>1</sup> |
|----------------------------|------------|------------|----------------------|
| Preferred Term | (N=xx) | (N=xx) | _ |
| - Any Adverse Events - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| SOC | | | |
| - Overall - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) | |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) | |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

<sup>&</sup>lt;sup>1</sup> Fisher's exact test

#### Table 91: Number and Percentage of Subjects with Adverse Events During Weeks 1 & 2

Same as Table 90 except only the first 2 weeks

#### Table 92: Number and Percentage of Subjects with Adverse Events During Weeks 3-12

Same as Table 90 except only the last 10 weeks

Table 93: Summary of Subjects with Adverse Events by Severity and Relationship – Oxytocin

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | M | ild | Mod | lerate | Sev | vere | Life-thr | eatening | | All Grades | |
| | MedDRA | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| SOC | PT | | | | | | | | | | | |
| | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 94: Summary of Subjects with Adverse Events by Severity and Relationship – Placebo

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | |
| SOC | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 95: Number and Percentage of Subjects with Adverse Events by Maximum Severity

| MedDRA SOC/ | | Pla | cebo | | Oxytocin | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | | (N=xx) | | | | (N= | =xx) | Т |
| | Mild | Moderate | Severe | Life-<br>threatening | Mild | Moderate | Severe | Life-<br>threatening |
| - Any Adverse Events - SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - Preferred term 1 | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) | nn (xx.x%)<br>nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 96: Number and Percentage of Subjects with Adverse Events by Maximum Severity During Weeks 1& 2

Same as Table 95 using only first 2 weeks

Table 97: Number and Percentage of Subjects with Adverse Events by Maximum Severity During Weeks 3-12

Same as Table 95 using only weeks 3-12

Table 98: Number and Percentage of Subjects with Adverse Events Occurring in >= 5%

| MedDRA SOC/ | Placebo | Oxytocin | |
|------------------|------------|------------|----------------------|
| Preferred Term | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| SOC | nn (xx.x%) | nn (xx.x%) | 0.xxx |
| - Overall - | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | 0.xxx |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | 0.xxx |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term. At least 5% occurring in either arm to be included in the table.

1 Fisher's Exact test

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 99: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study

| MedDRA SOC/ | Placebo | Oxytocin |
|------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| | | I |
| SOC | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 100: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Medication

| MedDRA SOC/ | Placebo | Oxytocin |
|------------------|------------|------------|
| Preferred Term | (N=xx) | (N=xx) |
| SOC | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | , , , |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

**Table 101:** CIWA-AR Score ≥ 10 at Least Once During Treatment

| | | | | | | | 95% | CI |
|---|---|---|---|---|---|---|---|---|
| | Placebo | Oxytocin | Total | | | | | |
| | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> | Cohen's h | Odds Ratio | OR Lower CI | OR Upper CI |
| CIWA-AR Score >= 10 | | | | | | | | |
| Never | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | | | | |
| At Least Once | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |

1 Chi-squared test

Table 102: Summary of Vital Signs and Body Weights

| Parameter | N | Mean | SD | Med | Max | Min |
|--------------------------------|----|------|------|------|------|------|
| Vital Sign (units) | | | | | | |
| Screening | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Oxytocin | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Week 1 | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Oxytocin | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Change from baseline | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Oxytocin | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Weeks 1, 2, 3, 4, 6, 8, 10, 13 | | | | | | |

Programmers note: vital signs include pulse rate, systolic blood pressure, and diastolic blood pressure. Body weight (lbs) will also be presented for screening, Weeks 6, 8, 10 and 13.

Table 103: Incidence of Abnormal Findings on Physical Exam in Nasal Mucosa

| | Placebo | Oxytocin |
|----------------------|------------|------------|
| | (N=xx) | (N=xx) |
| Abnomal Nasal Mucosa | nn (xx.x%) | nn (xx.x%) |

**Table 104:** Summary of Other Services Used During Treatment Period

| | Placebo | Oxytocin |
|--------------------|---------|----------|
| Services | (N=xx) | (N=xx) |
| Self Help Meetings | | |
| N | XX | XX |
| Mean | XX.X | XX.X |
| SD | XXX.XX | XXX.XX |
| Median | XX | XX |
| Min-Max | (xx-xx) | (xx-xx) |

| | Placebo | Oxytocin |
|---|---|---|
| Services | (N=xx) | (N=xx) |
| Have you visited another health professional to get help reducing drinking? | | |
| N | Xx | XX |
| Yes n (%) | xx (xx) | xx (xx) |

Programmer note: categorize type of professional for those categories reaching 5%

**Table 105:** Summary of ECG Results

| | ASP8062 | Placebo |
|--------------------------------------|------------|------------|
| Result | (N=xx) | (N=xx) |
| Screening | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| End of Study | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |

**Table 106:** Summary of Blood Chemistries

| | | Placebo | | | | Oxytocin | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Test | N | Mean | SD | Med | Min | Max | N | Mean | SD | Med | Min | Max |
| Test Name (units) | | | | | | | | | | | | |
| Screening | | | | | | | | | | | | |
| Week 6 | | | | | | | | | | | | |
| Change from baseline | | | | | | | | | | | | |
| Weeks 8, 10, 13 | | | | | | | | | | | | |

Programmers note: table will include creatinine, ALT, AST, total bilirubin, creatinine, sodium, and potassium.

Table 107: Summary of Positive Urine Drug Tests, Pregnancy Test or BAC > 0.000 Any Time During the Study

| | Number (% Positive) | |
|-----------------|---------------------|----------|
| Test | Placebo | Oxytocin |
| THC | xx (xx%) | xx (xx%) |
| Cocaine | xx (xx%) | xx (xx%) |
| Opioids | xx (xx%) | xx (xx%) |
| Methamphetamine | xx (xx%) | xx (xx%) |
| Amphetamine | xx (xx%) | xx (xx%) |
| Benzodiazapines | xx (xx%) | xx (xx%) |
| Buprenorphine | xx (xx%) | xx (xx%) |
| Methadone | xx (xx%) | xx (xx%) |
| Oxycodone | xx (xx%) | xx (xx%) |
| MDMA | xx (xx%) | xx (xx%) |
| Barbiturates | xx (xx%) | xx (xx%) |
| Pregnancy | xx (xx%) | xx (xx%) |
| BAC > 0.000 | xx (xx%) | xx (xx%) |

Table 108: BPAQ – Each Evaluation During Maintenance Period

| | | | 0 | xytocin | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Physical Aggression | | | | | | | | | | | | |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Verbal Aggress | ion | | | | | | | | | | | |

| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Hostility | | | | | | | | | | | | |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Anger | | | | | | | | | | | | |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 109: BPAQ Physical Aggression Score -- Full Model, Mixed Effects, Entire Maintenance Period

Type III Wald Tests<sup>1</sup>

| Parameter | Num DF | Den DF | F Value | p-value |
|-------------------------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Baseline<br>Total Score | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Values in Type III table are based upon transformed data {note to specify which transformation}

#### **Least Squares Means**

| | | | | 95% | 95% CI | | | Untran | sformed | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 10 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | 13 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 13 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 110: BPAQ Verbal Aggression Score -- Full Model, Mixed Effects, Entire Maintenance Period

Shell is same style as Table 109

Table 111: BPAQ Anger Score -- Full Model, Mixed Effects, Entire Maintenance Period

Shell is same style as Table 109

Table 112: BPAQ Hostility Score -- Full Model, Mixed Effects, Entire Maintenance Period

Shell is same style as Table 109

Table 113: SNAQ – Untransformed, Each Evaluation During Maintenance Period

| | | Oxytocin | | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

**Table 114:** SNAQ Score ≤ 14 at Each Visit During Treatment

| | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|
| | Placebo | Oxytocin | Total | | | | | |
| | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> | Cohen's h | Odds Ratio | OR Lower CI | OR Upper CI |
| SNAQ Score ≤ 14 | | | | | | | | |
| Week 6 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |
| Week 8 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |
| Week 10 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |
| Week 13 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |

1 Chi-squared test

Table 115: SNAQ Total Score -- Full Model, Mixed Effects, Entire Maintenance Period

Shell is same style as Table 109

Table 116: Frequency of Subjects with Suicidal Ideation Any Time During the Study

| Number of Subjects Re | Number of Subjects Reporting Suicidal Ideation by C-SSRS (%) | |
|---|---|---|
| Placebo Oxytocin p-value | | |
| (N=xx) | (N=xx) | |
| xx (xx.x%) | xx (xx.x%) | 0.xxx |

## 12.1.5 Exploratory Analyses

**Table 117:** Moderator: MINI AUD (Percent Heavy Drinking Days Weeks 3-12)

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|----------------------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 11 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Baseline<br>MINI AUD | 1 | XXX | XXX.XX | 0.xxx |
| ARM*MINI<br>AUD | 1 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | Louis Se uni es ivients | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | | | |
| AUD Split | Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| Yes | Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | xx.xxx |
| | Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| No | Oxytocin | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | xx.xxx |
| | Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

**Table 118:** Moderator: POMS Tension-Anxiety (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

**Table 119:** Moderator: POMS Depression-Dejection (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

Table 120: Moderator: ECR-RS Attachment-Related Anxiety (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

**Table 121:** Moderator: STAI (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

**Table 122:** Moderator: Drinking Goal (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

**Table 123:** Moderator: BIS Self Control (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

Table 124: Moderator: BIS Impulsive Behavior (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

**Table 125:** Moderator: Hyperkatifeia (Percent Heavy Drinking Days Weeks 3-12)

Shell style similar to Table 117

 Table 126:
 Hyperkatifeia Total Score

| | | Oxytocin | | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| Baseline | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 127: Hyperkatifeia Total Score- Generalized Linear Model, Week 13

## **Type III Wald Tests**

| Parameter | Num DF | Den DF | F Value | p-value |
|---------------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Hyperkatifeia | 1 | XXX | XXX.XX | 0.xxx |

## **Least Squares Means**

100

| | | | 95% CI | | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Oxytocin | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | xx.xxx | 0.xxx | XX.XXX |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 128: Hyperkatifeia Stress/Anxiety Score

Same as Table 126

Table 129: Hyperkatifeia Stress/Anxiety Score- Generalized Linear Model, Week 13

Same as Table 127

Table 130: Hyperkatifeia Depression Score

Same as Table 126

Table 131: Hyperkatifeia Depression Score- Generalized Linear Model, Week 13

Same as Table 127

**Table 132:** Hyperkatifeia Irritable Score

Same as Table 126

Table 133: Hyperkatifeia Irritable Score- Generalized Linear Model, Week 13

Same as Table 127

Table 134: Hyperkatifeia Pain Score

Same as Table 126

Table 135: Hyperkatifeia Pain Score- Generalized Linear Model, Week 13

## 12.2 Listings

**Listing 1:** Subject Disposition - All Subjects

| Subject<br>ID | Date of<br>Consent | Treatment<br>Group | Full<br>Analysis<br>Set | Study<br>Completi<br>on | (Day) Date of<br>Study Completion<br>or Early<br>Discontinuation | Reason for Early<br>Discontinuation | Subject<br>confined<br>or incar-<br>cerated | Start Date/ End<br>Date of<br>confinement |
|---|---|---|---|---|---|---|---|---|
| xxx | mm/dd/yyyy | Oxytocin | Yes | Yes | (xx) mm/dd/yyyy | xxxxxx | Yes | mm/dd/yyyy /<br>mm/dd/yyyy |
| | | Placebo | No | No | | | No | |
| | | None | | | | | | |

Note: Day is relative to Study Day 0.

**Listing 2:** Enrollment and Randomization – All Consented Subjects

| Subject<br>ID | Treatment<br>Group | Date of<br>Consent | Did the subject meet all eligibility criteria? | Randomized? | Date of<br>Randomization | Kit<br>Number |
|---|---|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Yes | Yes | mm/dd/yyyy | XXX |
| | Placebo | | No | No | | |

103

**Listing 3:** Reason not Eligible – Screen Failures

| Subject ID | Criterion Type | Criterion |
|------------|--------------------|-----------|
| XXX | Inclusion Criteria | |
| | Exclusion Criteria | |

**Listing 4:** Protocol Deviations

| Subject<br>ID | Treatment<br>Group | Deviation<br>Date | Protocol Deviation | Details |
|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Subject Failed to Meet the Inclusion/Exclusion Criteria | |
| AAA | Placebo | mini da, y y y y | Source Documentation was Not Available | |
| | | | Pregnancy Test Not Performed | |
| | | | Required study data was not obtained or obtained late due to site error | |
| | | | Informed Consent Deviation | |
| | | | AE/SAE Reporting Deviation | |
| | | | Other Deviation: | xxxxxxxxxxxx |

104

Note: Only subjects with protocol deviation are listed.

**Listing 5:** Subjects Excluded from the Efficacy Analysis

| Subject<br>ID | Treatment<br>Group | Reason for Exclusion from FA |
|---------------|---------------------|------------------------------|
| Xxx | Overtagin | |
| AXX | Oxytocin<br>Placebo | XXXXXX |

Note: Only subjects excluded from the efficacy analysis are listed.

**Listing 6:** Demographics Data

| Subject<br>ID | Treatment<br>Group | Gender | Age<br>(yrs) | Ethnicity | Race | Marital Status |
|---|---|---|---|---|---|---|
| XXX | Oxytocin | Male | XX | Hispanic or Latino | American Indian or Alaska Native | Married |
| | | | | Not Hispanic or | | |
| | Placebo | Female | | Latino | Asian | Divorced |
| | | | | Unknown | Native Hawaiian or Other Pacific Islander | Living with Partner |
| | | | | | Black or African American | Widowed |
| | | | | | White | Separated |
| | | | | | Other | Never Married |
| | | | | | Unknown | Unknown |
| | | | | | | Missing |

| Subject<br>ID | Treatment<br>Group | Years of Education | Years of Formal Education (GED=12years) | Usual Employment Pattern in the last 30 days |
|---|---|---|---|---|
| XXX | Oxytocin | XX | XXX | Full-time, 35+ hrs/week |
| | Placebo | | | Part-time, regular hours |
| | | | | Part-time, irregular |
| | | | | hours/daywork |
| | | | | Student |
| | | | | Military service |
| | | | | Unemployed |
| | | | | Retired/Disabled |
| | | | | Homemaker |
| | | | | In controlled environment |
| | | | | Unknown |
| | | | | Unknown |

**Listing 7:** Baseline Drinking Characteristics

| Subject | Treatment | Drinks/Week | Drinks/Week<br>(Days -1 to -7<br>Pre- | % Change<br>Drinks per<br>Week Pre-<br>screen to Pre- | Drinks/<br>Drinking Day | Drinks/Drinking<br>Day (Days -1 to -<br>7 Pre- | % Change<br>DPDD Pre-<br>screen to Pre- |
|---|---|---|---|---|---|---|---|
| ID ° | Group | (Days -1 to -28) | randomization) | randomization | (Days -1 to -28) | randomization) | randomization |
| XXX | Oxytocin | XXX.X | XXX.X | XX.X | XXX.X | XXX.X | XX.X |
| | Placebo | | | | | | |

| Subject<br>ID | Treatment<br>Group | Weekly % Heavy<br>Drinking Days<br>(Days -1 to -28) | Weekly % Days<br>Abstinent<br>(Days -1 to -28) | WHO Risk<br>Level |
|---|---|---|---|---|
| XXX | Oxytocin | XXX.X | XXX.X | High Risk |
| | Placebo | | | Very High Risk |

**Listing 8: MINI DSM5 Disorders** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Diagnosis | Timeframe |
|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | xxxxxx | Current (2 weeks) |
| | Placebo | | | Past |
| | | | | Recurrent |

Note: Only subjects with a diagnosis of a disorder will be listed.

**Listing 9:** MINI DSM5 AUD

| Subject<br>ID | Treatment<br>Group | Visit Date | # of Symptoms |
|---------------|--------------------|------------|---------------|
| VVV | Oxytocin | mm/dd/yyyy | VV |
| XXX | Placebo | mm/dd/yyyy | XX |
Listing 10: MINI AUD End of Study

| Subject<br>ID | Treatment<br>Group | | | | | | Item | | | | | | # of Symptoms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| XXX | Oxytocin | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | |
| | Placebo | N | N | N | N | N | N | N | N | N | N | N | |
| | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |

| Item # | List of Items |
|---|---|
| 1 | a. During the times when you drank alcohol, did you end up drinking more than you planned when you started? |
| 2 | b. Did you repeatedly want to reduce or control your alcohol use? Did you try to cut down or control your alcohol use, but failed? IF YES TO EITHER, MARK YES. |
| 3 | c. On the days that you drank, did you spend substantial time obtaining alcohol, drinking, or recovering from the effects of alcohol? |
| 4 | d. Did you crave or have a strong desire or urge to use alcohol? |
| 5 | e. Did you spend less time meeting your responsibilities at work, at school, or at home, because of your repeated drinking? |
| 6 | f. If your drinking caused problems with your family or other people, did you still keep on drinking? |
| 7 | g. Were you intoxicated more than once in any situation where you or others were physically at risk, for example, driving a car, riding a motorbike, using machinery, boating, etc.? |
| 8 | h. Did you continue to use alcohol, even though it was clear that the alcohol had caused or worsened psychological or physical problems? |
| 9 | i. Did you reduce or give up important work, social or recreational activities because of your drinking? |
| 10 | j. Did you need to drink a lot more in order to get the same effect that you got when you first started drinking or did you get much less effect with continued use of the same amount? |
| 11 | K1. When you cut down on heavy or prolonged drinking did you have any of the following: [increased sweating or heart rate; hand tremor or "the shakes"; trouble sleeping; nausea or vomiting; hearing or seeing things other people could not see or hear or having sensations in your skin for no apparent reason; agitation; anxiety; seizures] (If yes to 2 or more of these, check yes for this question), OR K2. Did you drink alcohol to reduce or avoid withdrawal symptoms or to avoid being hung over? If K1 or K2 = yes, then score as yes. |

**Listing 11: Medical History** 

| Subject<br>ID No. | Treatment<br>Group | SOC | Specify (Preferred Term/<br>Verbatim Term) | Start Date | Ongoing |
|---|---|---|---|---|---|
| | • | | | | 9 9 |
| | | Blood and Lymphatic System | | | |
| XXX | Oxytocin | Disorders | Xxxxxxxxxx/ xxxxxxxx | mm/dd/yyyy | No |
| | Placebo | Cardiac Disorders | | | Yes |
| | | Congenital, Familial and Genetic Disorders | | | |
| | | Ear and Labyrinth Disorders | | | |
| | | Endocrine Disorders | | | |
| | | Eye Disorders | | | |
| | | Gastrointestinal Disorders | | | |
| | | General Disorders and<br>Administration Site Conditions | | | |
| | | Hepatobiliary Disorders | | | |
| | | Immune System Disorders | | | |
| | | Infections and Infestations | | | |
| | | Injury, Poisoning and Procedural Complications | | | |
| | | Investigations | | | |
| | | Metabolism and Nutrition Disorders | | | |
| | | Musculoskeletal and Connective<br>Tissue Disorders | | | |
| | | Neoplasms Benign, Malignant<br>and Unspecified (incl Cysts and<br>Polyps) | | | |
| | | Nervous system Disorders | | | |
| | | Pregnancy, Puerperium and<br>Perinatal Conditions | | | |
| | | Psychiatric Disorders | | | |

| Renal and Urinary Disorders |
|---------------------------------|
| Reproductive System and Breast |
| Disorders |
| Respiratory, Thoracic and |
| Mediastinal Disorders |
| Skin and Subcutaneous Tissue |
| Disorders |
| Social Circumstances |
| Surgical and Medical Procedures |
| Vascular Disorders |
| Other:xxxxxxxx |

**Listing 12:** Surgical History

| Subject<br>ID No. | Treatment<br>Group | Has the subject had any past surgeries? | Date of Surgery | Type of Surgery |
|---|---|---|---|---|
| XXX | Oxytocin | Yes | mm/dd/yyyy | XXXXXXXXXXX |
| • | Placebo | No | | |

**Listing 13:** Physical Exam

| Subject<br>ID No. | Treatment<br>Group | Exam Date | Any abnormal finding during the physical exam? | Describe |
|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Yes | XXXXXXX |
| | Placebo | | No | |

Programming Note: Only report the items that are abnormal

**Listing 14:** Drinking Treatment History

| Subject<br>ID No. | Treatment<br>Group | Age first<br>started<br>drinking<br>alcohol<br>regularly | Number of lifetime inpatient visits to get help with reducing or quitting drinking | Number of lifetime inpatient hospitalizations for illnesses, injuries, or accidents due to drinking | Number of times in lifetime underwent alcohol detoxification using medication | Number of lifetime outpatient visits with a health professional to get help with reducing or quitting drinking | Number of group<br>meetings<br>attended for<br>alcohol problems<br>or drinking in<br>the past year |
|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | | | | | | |

Listing 15: Drinking Goal

| | | | | Subjects wanting to reduce drinking, expected drinks per day | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Which treatment goal would you like to achieve by the end of the study? | | Mon | Tues | Wed | Thur | Fri | Sat | Sun |
| XXX | Oxytocin | mm/dd/yyyy | Abstinence | X | X | X | X | X | X | х |
| | Placebo | | Reduction but not stop | | | | | | | |

| Subject<br>ID | Treatment<br>Group | Visit Date | How motivated to reach your goal? | How confident to achieve your goal? |
|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | 1=Not Motivated | 1=Not Confident |
| | Placebo | | 2, 3, 4, 5, 6, 7, 8, 9 | 2, 3, 4, 5, 6, 7, 8, 9 |
| | | | 10=Extremely Motivated | 10=Extremely Confident |
| | | | Refuse to answer | Refuse to answer |

Listing 16: Daily and Weekly Standard Drink Units (TLFB) During Treatment

| Subject<br>ID | Treatment<br>Group | Week | D1 | D2 | D3 | <b>D</b> 4 | D5 | D6 | <b>D</b> 7 | Mean<br>drinks/day | Mean drinks/<br>drinking day | Heavy<br>drinking days | % days<br>abstinent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | 1 | XX | XX | XX | XX | XX | XX | XX | XX.XX | XX.XX | XX.XX | XX |
| | Placebo | 2 | | | | | | | | | | | |
| | | 3, etc | | | | | | | | | | | |

**Listing 17: Drinking Question** 

| Subject<br>ID | Treatment<br>Group | Date of<br>Assessment | Did the subject have any drinking days since the last visit? | Did the subject have any heavy drinking days since the last visit? | Date of last visit |
|---|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Yes | Yes | mm/dd/yyyy |
| | Placebo | | No | No | |
| • | | | | | |

Listing 18: Drinking Consequences, Craving, Appetite, and Anxiety

| Subject<br>ID | Treatment<br>Group | Week | Urge to Drink | CIWA-AR | STAI | SNAQ | ECR-RS<br>Attachment-<br>Related Anxiety | BIS Total Score |
|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | XX | | XX | XX | XX | XX | XX |
| | Placebo | | | | | | | |

**Listing 19: UPSIT Scores** 

| Subject<br>ID | Treatment<br>Group | Week | Total Score | Category |
|---------------|--------------------|------|-------------|--------------------|
| XXX | Oxytocin | XX | XX | Normosmia |
| | Placebo | | | Mild microsmia |
| | | | | Moderate microsmia |
| | | | | Severe microsmia |
| | | | | Anosmia |
| | | | | Normosmia |

**Listing 20:** POMS Scores

| Subject<br>ID | | | Scores | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment<br>Group | Week | Total Mood<br>Disturbance | Tension | Depression | Anger | Fatigue | Confusion | Vigor |
| XXX | Oxytocin | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | | | | | | | | |

**Listing 21: PROMIS Scale Scores** 

| Subject<br>ID | Treatment<br>Group | Week | Sleep Disturbance | Alcohol Negative<br>Consequences | Pain Interference |
|---|---|---|---|---|---|
| XXX | Oxytocin | XX | XX | xx | XX |
| | Placebo | | | | |

**Listing 22:** Smoking Data

| Subject<br>ID | Treatment<br>Group | Week | Visit Date | Over the past week, how many days did you smoke cigarettes? | On the days you smoked, how many cigarettes did you smoke on average? | How many days did you use other tobacco or nicotine products during the past week? |
|---|---|---|---|---|---|---|
| XXX | Oxytocin | 1, 6, 8, 10, 13 | mm/dd/yyyy | x | XX | X |
| | Placebo | 1, 0, 0, 10, 13 | | | | |

**Listing 23:** Exit Interview

| Subject<br>ID | Treatment<br>Group | Visit Date | What study drug do<br>you believe you<br>were taking? | Why do you think you received that drug? | Do you feel the study drug helped you to reduced drinking? | How would you describe your experience taking the study drug? |
|---|---|---|---|---|---|---|
| xxx | Oxytocin | mm/dd/yyyy | Placebo | Had side effects | Very Much | Experienced no unwanted side effects and benefited from taking the medication |
| | Placebo | | Active medication | Had no side effects | Much | Experienced some unwanted side effects but benefited from taking the medication |
| | | | Both placebo and active | Staff told me | Moderately | Experienced a lot unwanted side effects but benefited from taking the medication |
| | | | Don't know | Staff treatment me different | A Little | Experienced no unwanted side effects but did not benefit from taking the medication |
| | | | Other substance | No improvement in drinking | Not Little | Experienced some unwanted side effects and did not benefit from taking the medication |
| | | | | Had improvement in drinking | Not at all | Experienced a lot of unwanted side effects and did not benefit from taking the medication |
| | | | | Had a hunch | | |
| | | | | I just felt different | | |
| | | | | Other: xxxxx | | |

| Subject<br>ID | Treatment<br>Group | Visit Date | If a friend were in need of help<br>for a drinking problem, would<br>you recommend taking the study<br>drug to him/her? | If you were to need treatment in the future, would you choose to take the study drug again? | How much do you think of yourself as wanting to please other people (people pleaser)? |
|---|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Yes, definitely | Definitely yes | More than average |
| | Placebo | | Yes, generally | Probably yes | Average |
| | | | Neither yes nor no | Maybe | Less than average |
| | | | No, not really | Probably not | |
| | | | No, definitely not | Definitely not | |

**Listing 24:** Other Services Use

| Subject<br>ID | Group | Date | Week | Since your last visit<br>did you attend any<br>AA, 12-step, SOS, or<br>similar group<br>meeting? | How many? | Have you visited another health professional to get help reducing drinking? | What type of professional? |
|---|---|---|---|---|---|---|---|
| XXX | Oxytocin<br>Placebo | mm/dd/yyyy | XX | Yes<br>No | XXXX | Yes<br>No | XXXXX |

**Listing 25:** Drug Exposure

| Subject<br>ID No. | Treatment<br>Group | Study<br>Month | Date Start of<br>Month | Date End of<br>End of<br>Month | Volume of<br>Drug<br>Prescribed | Volume of<br>Drug<br>Taken | Reason for Discontinuation |
|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | 1, 2, 3 | mm/dd/yyyy | mm/dd/yyyy | xx | XX | |
| | Placebo | | | | | | |

**Listing 26:** Adverse Events

| Subject<br>ID | Treatment<br>Group | Adverse Event (Verbatim) S: SOC P: PT Term | Start Date/<br>Day | Stop Date/<br>Day | Duration<br>in Days | Severity | Relation<br>-ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | Verbatim | mm/dd/yyyy | mm/dd/yyyy | | 1 | 1 | 1 | 1 | Yes |
| | Placebo | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

**Listing 27:** Adverse Events Leading to Subject Discontinuation from Study

| Subject<br>ID | Treatment<br>Group | Adverse<br>Event<br>(Verbatim)<br>S: SOC<br>P: PT<br>Term | Start Date/<br>Day | Stop Date/<br>Day | Duration in Days | Severity | Relation<br>-ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | Verbatim | mm/dd/yyyy | mm/dd/yyyy | | 1 | 1 | 1 | 1 | Yes |
| | Placebo | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

Listing 28: Adverse Events Leading to Discontinuation of Investigational Product

| Subject<br>ID | Treatment<br>Group | Adverse Event (Verbatim) S: SOC P: PT Term | Start Date/<br>Day | Stop Date/<br>Day | Duration in Days | Severity | Relation<br>-ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | Verbatim | mm/dd/yyyy | mm/dd/yyyy | | 1 | 1 | 1 | 1 | Yes |
| | Placebo | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

**Listing 29: Serious Adverse Events** 

| Subject<br>ID | Treatment<br>Group | SAE<br>Verbatim<br>S: SOC<br>P: PT | Start Date/<br>Day | Stop Date/<br>Day | SAE Category | Severity | Relationship |
|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | Verbatim | mm/dd/yyyy | mm/dd/yyyy | Death | 1 | 1 |
| | Placebo | S: XXX | Xx | Xx | Life-threatening | 2 | 2 |
| | | P: XX | | | Hospitalization | 3 | 3 |
| | | | | | Disability | 4 | 4 |
| | | | | | Congenital Anomaly/Birth<br>Defect | 5 | 5 |
| | | | | | Required Intervention to Prevent<br>Permanent Impairment / Damage | | |
| | | | | | Other | | |

| Subject<br>ID No. | SAE | Continued<br>Study<br>Participation | Study Drug<br>Start Date | Date of last<br>administration<br>of study drug<br>prior to SAE | SAE Abated<br>after study<br>drug<br>stopped? | Continued study drug Administration | SAE<br>reappeared<br>after<br>rechallenge? | Outcome |
|---|---|---|---|---|---|---|---|---|
| XXX | Verbatim | Yes | mm/dd/yyyy | mm/dd/yyyy | Yes | Yes | Yes | 1 |
| | | No | | | No | No | No | 2 |
| | | | | | n/a | | n/a | 3 |

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Outcome: 1=Recovered/Resolved; 2=Recovering/Resolving; 3=Not Recovered/Not Resolved; 4=Recovered/Resolved With Sequelae; 5=Fatal (Date of Death)

**Listing 30:** Columbia-Suicide Severity Scale

| | | | | Response to Question: | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjec<br>t ID | Treatment<br>Group | Visit Date | Study<br>Week | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q13 |
| XXX | Oxytocin | mm/dd/yyyy | 1, 2, 5 | Yes | Yes | Yes | Yes | Yes | Yes | Type 1 | 1 | 1 | 0 | 0 | 0 | Yes |
| | Placebo | | 9, 13 | No | No | No | No | No | No | Type 2 | 2 | 2 | 1 | 1 | 1 | No |
| | | | | | | | | | | Type 3 | 3 | 3 | 2 | 2 | 2 | |
| | | | | | | | | | | Type 4 | 4 | 4 | 3 | 3 | 3 | |
| | | | | | | | | | | Type 5 | 5 | 5 | 4 | 4 | 4 | |
| | | | | | | | | | | | | | 5 | 5 | 5 | |

#### **Suicide Ideation**

- 1. Have you wished you were dead or wished you could go to sleep and not wake up?
- 2. Have you actually had any thoughts of killing yourself?
- 3. Have you been thinking about how you might do this?
- 4. Have you had these thoughts and had some intention of acting on them?
- 5. Have you started to work out or worked out the details of how to kill yourself?
- 6. Do you intend to carry out this plan?

#### **Intensity of Ideation**

- 7. The following features should be rated with respect to the most severe type of ideation (i.e. 1-5 with 1 being the least severe and 5 being the most severe)
- 8. How many times have you had these thoughts?1=Less than once a week; 2=Once a week; 3=2-5 times a week; 4=Daily or almost; 5=Many times each day
- 9. When you have the thoughts, how long do they last? 1=Fleeting-few seconds or minutes; 2=Less than 1 hr-some of the time; 3=1-4 hrs/a lot of time; 4=4-8 hrs/most of day; 5=More than 8 hours/persistent or continuous
- 10. Could/can you stop thinking about killing yourself or wanting to die if you want to? 1=Easily; 2=Little Difficulty; 3=Some Difficulty; 4=Lot of Difficulty; 5=Unable to control; 0=Does not attempt to control
- 11. Are there things that stop you from wanting to die or acting on thoughts of committing suicide? 1=Definite deterrents; 2=Probably Deterrents; 3=Uncertain Deterrents; 4=Unlikely Deterrents; 5=No Deterrents; 0=Does not apply
- 12. What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end pain or stop the way you were feeling or to get attention, revenge or reaction from others 1=Completely to get attention or revenge or reaction; 2=Mostly to get attention or revenge or reaction; 3=Equally to get attention or revenge or reaction and stop pain; 4=Mostly to stop pain; 5=Completely to stop pain; 0=Does not apply

#### **Suicidal Behavior**

- 13. Have you made a suicide attempt?
- 14. Number of attempts
- 15. Has the subject engaged in non-suicidal self-injurious behavior?
- 16. Has there been a time when you started to do something to end your life but someone or something stopped you before actually did anything?
- 17. Number interrupted
- 18. Has there been a time when you stared to do something to try to end your life but you stopped yourself before you actually did anything?
- 19. Number aborted
- 20. Have you taken any step towards making a suicide attempt or preparing to kill yourself?
- 21. Suicidal behavior was present during the assessment period
- 22. Completed suicide?
- 23. Actual Lethality/Medical Damage; 0=No physical damage; 1=Minor physical damage; 2=Moderate physical Damage; 3=Moderately severe physical damage; 4=Severe physical damage; 5=Death
- 24. Potential Lethality; 0=Behavior not likely to result in injury; 1=Behavior likely to result in injury, but not death; 2=Behavior likely to result in death

Listing 31: BPAQ Scores

| | | | | Scores | | |
|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Week | Physical<br>Aggression | Verbal<br>Aggression | Hostility | Anger |
| XXX | Oxytocin | XX | XXX | XXX | XXX | XXX |
| | Placebo | | | | | |

**Listing 32:** Blood Chemistries

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result | Units | Flag | Evaluation |
|---|---|---|---|---|---|---|---|
| xxxx | Oxytocin | mm/dd/yyyy | Creatinine | X.XX | mg/dL | H (high) | WNL |
| | Placebo | | Total Bilirubin | XXX | mg/dL | L (low) | Abnormal, NCS |
| | | | ALT | XX.X | U/L | | Abnormal, CS |
| | | | AST | X.XX | U/L | | |
| | | | sodium | XX.X | U/L | | |
| | | | Potassium | | | | |

**Listing 33: Pregnancy Test/Birth Control Data** 

| Subject ID | Treatment Group | Pregnancy Test<br>Performed? | Pregnancy Test<br>Date | Pregnancy<br>Result | Methods of birth control |
|---|---|---|---|---|---|
| XXX | Oxytocin | Not Done | mm/dd/yyyy | Negative | Oral Contraceptive |
| | Placebo | | | Positive | Contraceptive Sponge |
| | | | | | Contraceptive Skin Patch |
| | | | | | Double Barrier |
| | | | | | Intrauterine |
| | | | | | Etonogestrel implant |
| | | | | | Medroxyprogesterone |
| | | | | | Complete Abstinence |
| | | | | | Hormonal Vaginal contraceptive Ring |
| | | | | | Surgically Sterile |
| | | | | | Postmenopausal |
| | | | | | Partner surgically Sterile |
| | | | | | Other: xxxxxxxxxxxxxx |

Programming note: Only indicate birth control methods that were indicated as Yes

Listing 34: **Blood Alcohol Concentration** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | BAC<br>Performed | Time of BAC | BAC % |
|---|---|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Screen | Done | hh:mm | x.xxx |
| | Placebo | | 1, 2, 3 | Not Done | | |
| | | | 4, 6, 8 | | | |
| | | | 10, 13 | | | |

**Listing 35:** Urine Drug Screen

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | AMP<br>a,b | Benzos | Barb | Coc | Bup | EGT | MDMA | Meth | Methadone | Opioids | Оху | THC |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | mm/dd/yyyy | Screen | P | P | P | P | P | P | P | P | P | P | P | P |
| | Placebo | | 1, 2, 3 | N | N | N | N | N | N | N | N | N | N | N | N |
| | | | 4, 6, 8 | | | | | | | | | | | | |
| | | | 10, 13 | | | | | | | | | | | | |

 <sup>&</sup>lt;sup>a</sup> P=positive; N=negative
 <sup>b</sup> AMP=amphetamine, Benzos=benzodiazepines, Coc=cocaine, Meth=methamphetamine, Oxy=oxycodone, Bup=buprenorphine, Barb=barbiturates

**Listing 36:** Vital Signs and Body Weights

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | Weight (Kg) | Heart Rate<br>(beats/min) | Systolic Pressure (mmHg) | Diastolic Pressure<br>(mmHg) |
|---|---|---|---|---|---|---|---|
| | | /11/ | G : | | | | |
| XXX | Oxytocin | mm/dd/yyyy | Screening | XXX | XXX | XXX | XXX |
| | Placebo | | 4 | | | | |
| | | | 8 | | | | |
| | | | 12, 16, 20 | | | | |
| | | | 24, 26, 27 | | | | |

**Listing 37: Prior and Concomitant Medications** 

| Subject<br>ID | Treatment<br>Group | Prior<br>Med? | Verbatim Med | Indication | Route | Frequency | Dose | Start Date | Stop Date | Continuing? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | Oxytocin | Yes | XXX | xxxxxx | XXXXXX | XXXXXX | XXXXXX | dd/mmm/yyyy | dd/mmm/yyyy | Yes |
| xxx | Placebo | No | XXX | | | | | | | No |

# 12.3 Figures

Figure 1: Percent Heavy Drinking Days per Week Least Squares Means – Untransformed



Programmer note: connect the week estimates for each treatment group using linear line join, 95% CI at each estimate, add Cohen's d to each point and \*p-value < 0.05

Figure 2: Mean Drinks per Week Least Squares Means – Untransformed

Shell style similar to Figure 1

Figure 3: Mean Drinks per Drinking Day by Week Least Squares Means – Untransformed

Shell style similar to Figure 1



Figure 4: Percentage of Subjects No Heavy Drinking Days Weeks 3-12

Programmer note: Use percent on y-axis, bar graph of PSNHDD add Cohen's h, \*a significant p-value, put values on graph and the programmer note is a significant p-value of the programmer note.

Figure 5: Percentage of Subjects Abstinent Weeks 3-12

Shell style similar to Figure 4

Oxytocin

Figure 6: Percentage of Subjects with WHO 1-Level Decrease in Alcohol Consumption Weeks 3-12
Shell style similar to Figure 4

Figure 7: Percentage of Subjects with WHO 2-Level Decrease in Alcohol Consumption Weeks 3-12

Statistical Analysis Plan: Protocol NCIG-007R, Version 1.0 Dated: 7 Sep 2023

**Placebo** 

Shell style similar to Figure 4

# Figure 8: Cumulative Grace Periods for Percentage of Subjects No Heavy Drinking Days

Shell style similar to Figure 4

Programmer note put all of the grace periods (full treatment period, 1 month, 2 months) on the same graph

# Figure 9: Cumulative Grace Periods for Percentage of Subjects Abstinent

Shell style similar to Figure 4

### Figure 10: Cumulative Grace Periods for Percentage WHO 1-Level Decrease in Alcohol Consumption

Shell style similar to Figure 4

### Figure 11: Cumulative Grace Periods for Percentage WHO 2-Level Decrease in Alcohol Consumption

Shell style similar to Figure 4



Figure 12: Percentage Days Abstinent per Week Least Squares Means – Untransformed

Programmer note: connect the week estimates for each treatment group using linear line join, add Cohen's d to each point and \*p-value <0.05

Figure 13: Weekly Number of Cigarettes Smoked in Smokers Least Squares Means – Untransformed Shell style similar to Figure 12

Figure 14: POMS Total Score Least Squares Means by Visit – Untransformed
Shell style similar to Figure 12

Figure 15: POMS Tension-Anxiety Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 16: POMS Depression-Dejection Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 17: POMS Vigor-Activity Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 18: POMS Fatigue-Inertia Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 19: POMS Anger-Hostility Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 20: POMS Confusion-Bewilderment Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 21: PROMIS Alcohol Negative Consequences Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 22: PROMIS Sleep Disturbances Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 23: PROMIS Pain Interference Least Squares Means by Visit – Untransformed

Shell style similar to Figure 12

Figure 24: ECR-RS Attachment-Related Anxiety Least Squares Means by Visit – Untransformed

134

Statistical Analysis Plan: Protocol NCIG-007R, Version 1.0 Dated: 7 Sep 2023

Shell style similar to Figure 12

Figure 25: Clinical Chemistry Values Over Time